CLINICAL TRIAL: NCT01763866
Title: A Double-blind, Randomized, Placebo and Ezetimibe Controlled, Multicenter Study to Evaluate Safety, Tolerability and Efficacy of AMG 145 on LDL-C in Combination With Statin Therapy in Subjects With Primary Hypercholesterolemia and Mixed Dyslipidemia
Brief Title: LDL-C Assessment With PCSK9 Monoclonal Antibody Inhibition Combined With Statin Therapy-2
Acronym: LAPLACE-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20110115; 2012-001363-70 (EudraCT Number)
Record Dates: First submitted 2013-01-07; First posted 2013-01-09 (Estimated); Results first posted 2015-12-22 (Estimated); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Hyperlipidemia
Keywords: High cholesterol, Treatment for high cholesterol, Lowering cholesterol, Lowering high cholesterol, Hypercholesterolemia
MeSH Terms: conditions — Hyperlipidemias; Hypercholesterolemia | interventions — evolocumab; Ezetimibe; Atorvastatin; Rosuvastatin Calcium; Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (24):
- A10 PBO Q2W (Placebo Comparator): Participants received atorvastatin 10 mg once daily during the 4 week lipid stabilization period and then in combination with placebo (PBO) subcutaneous injection once every 2 weeks (Q2W) and placebo tablets once daily for up to 12 weeks.
  Interventions: Drug: Placebo to Evolocumab; Drug: Placebo to Ezetimibe; Drug: Atorvastatin
- A10 PBO QM (Placebo Comparator): Participants received atorvastatin 10 mg a day during the 4-week lipid stabilization period and then with placebo subcutaneous injection once every month (QM) and placebo tablets once a day for up to 12 weeks.
  Interventions: Drug: Placebo to Evolocumab; Drug: Placebo to Ezetimibe; Drug: Atorvastatin
- A10 EZE (Q2W) (Active Comparator): Participants received atorvastatin 10 mg a day during the 4-week lipid stabilization period and then with placebo subcutaneous injection once every 2 weeks and 10 mg ezetimibe (EZE) orally once a day for up to 12 weeks.
  Interventions: Drug: Ezetimibe; Drug: Placebo to Evolocumab; Drug: Atorvastatin
- A10 EZE (QM) (Active Comparator): Participants received atorvastatin 10 mg a day during the 4-week lipid stabilization period and then with placebo subcutaneous injection once a month and 10 mg ezetimibe orally once a day for up to 12 weeks.
  Interventions: Drug: Ezetimibe; Drug: Placebo to Evolocumab; Drug: Atorvastatin
- A10 EvoMab Q2W (Experimental): Participants received atorvastatin 10 mg a day during the 4-week lipid stabilization period and then with 140 mg evolocumab (EvoMab) by subcutaneous injection once every 2 weeks and placebo tablets once a day for up to 12 weeks.
  Interventions: Biological: Evolocumab; Drug: Placebo to Ezetimibe; Drug: Atorvastatin
- A10 EvoMab QM (Experimental): Participants received atorvastatin 10 mg a day during the 4-week lipid stabilization period and then with 420 mg evolocumab by subcutaneous injection once a month and placebo tablets once a day for up to 12 weeks
  Interventions: Biological: Evolocumab; Drug: Placebo to Ezetimibe; Drug: Atorvastatin
- A80 PBO Q2W (Placebo Comparator): Participants received atorvastatin 80 mg a day during the 4-week lipid stabilization period and then with placebo subcutaneous injection once every 2 weeks and placebo tablets once a day for up to 12 weeks.
  Interventions: Drug: Placebo to Evolocumab; Drug: Placebo to Ezetimibe; Drug: Atorvastatin
- A80 PBO QM (Placebo Comparator): Participants received atorvastatin 80 mg a day during the 4-week lipid stabilization period and then with placebo subcutaneous injection once every month and placebo tablets once a day for up to 12 weeks.
  Interventions: Drug: Placebo to Evolocumab; Drug: Placebo to Ezetimibe; Drug: Atorvastatin
- A80 EZE (Q2W) (Active Comparator): Participants received atorvastatin 80 mg a day during the 4-week lipid stabilization period and then with placebo subcutaneous injection once every 2 weeks and 10 mg ezetimibe orally once a day for up to 12 weeks.
  Interventions: Drug: Ezetimibe; Drug: Placebo to Evolocumab; Drug: Atorvastatin
- A80 EZE (QM) (Active Comparator): Participants received atorvastatin 80 mg a day during the 4-week lipid stabilization period and then with placebo subcutaneous injection once a month and 10 mg ezetimibe orally once a day for up to 12 weeks.
  Interventions: Drug: Ezetimibe; Drug: Placebo to Evolocumab; Drug: Atorvastatin
- A80 EvoMab Q2W (Experimental): Participants received atorvastatin 80 mg a day during the 4-week lipid stabilization period and then with 140 mg evolocumab by subcutaneous injection once every 2 weeks and placebo tablets once a day for up to 12 weeks.
  Interventions: Biological: Evolocumab; Drug: Placebo to Ezetimibe; Drug: Atorvastatin
- A80 EvoMab QM (Experimental): Participants received atorvastatin 80 mg a day during the 4-week lipid stabilization period and then with 420 mg evolocumab by subcutaneous injection once a month and placebo tablets once a day for up to 12 weeks.
  Interventions: Biological: Evolocumab; Drug: Placebo to Ezetimibe; Drug: Atorvastatin
- R5 PBO Q2W (Placebo Comparator): Participants received rosuvastatin 5 mg a day during the 4-week lipid stabilization period and then with placebo subcutaneous injection once every 2 weeks for up to 12 weeks.
  Interventions: Drug: Placebo to Evolocumab; Drug: Rosuvastatin
- R5 PBO QM (Placebo Comparator): Participants received rosuvastatin 5 mg a day during the 4-week lipid stabilization period and then with placebo subcutaneous injection once every month for up to 12 weeks.
  Interventions: Drug: Placebo to Evolocumab; Drug: Rosuvastatin
- R5 EvoMab Q2W (Experimental): Participants received rosuvastatin 5 mg a day during the 4-week lipid stabilization period and then with 140 mg evolocumab by subcutaneous injection once every 2 weeks for up to 12 weeks.
  Interventions: Biological: Evolocumab; Drug: Rosuvastatin
- R5 EvoMab QM (Experimental): Participants received rosuvastatin 5 mg a day during the 4-week lipid stabilization period and then with 420 mg evolocumab by subcutaneous injection once a month for up to 12 weeks.
  Interventions: Biological: Evolocumab; Drug: Rosuvastatin
- R40 PBO Q2W (Placebo Comparator): Participants received rosuvastatin 40 mg a day during the 4-week lipid stabilization period and then with placebo subcutaneous injection once every 2 weeks for up to 12 weeks.
  Interventions: Drug: Placebo to Evolocumab; Drug: Rosuvastatin
- R40 PBO QM (Placebo Comparator): Participants received rosuvastatin 40 mg a day during the 4-week lipid stabilization period and then with placebo subcutaneous injection once every month for up to 12 weeks.
  Interventions: Drug: Placebo to Evolocumab; Drug: Rosuvastatin
- R40 EvoMab Q2W (Experimental): Participants received rosuvastatin 40 mg a day during the 4-week lipid stabilization period and then with 140 mg evolocumab by subcutaneous injection once every 2 weeks for up to 12 weeks.
  Interventions: Biological: Evolocumab; Drug: Rosuvastatin
- R40 EvoMab QM (Experimental): Participants received rosuvastatin 40 mg a day during the 4-week lipid stabilization period and then with 420 mg evolocumab by subcutaneous injection once a month for up to 12 weeks.
  Interventions: Biological: Evolocumab; Drug: Rosuvastatin
- S40 PBO Q2W (Placebo Comparator): Participants received simvastatin 40 mg a day during the 4-week lipid stabilization period and then with placebo subcutaneous injection once every 2 weeks for up to 12 weeks.
  Interventions: Drug: Placebo to Evolocumab; Drug: Simvastatin
- S40 PBO QM (Placebo Comparator): Participants received simvastatin 40 mg a day during the 4-week lipid stabilization period and then with placebo subcutaneous injection once every month for up to 12 weeks.
  Interventions: Drug: Placebo to Evolocumab; Drug: Simvastatin
- S40 EvoMab Q2W (Experimental): Participants received simvastatin 40 mg a day during the 4-week lipid stabilization period and then with 140 mg evolocumab by subcutaneous injection once every 2 weeks for up to 12 weeks.
  Interventions: Biological: Evolocumab; Drug: Simvastatin
- S40 EvoMab QM (Experimental): Participants received simvastatin 40 mg a day during the 4-week lipid stabilization period and then with 420 mg evolocumab by subcutaneous injection once a month for up to 12 weeks.
  Interventions: Biological: Evolocumab; Drug: Simvastatin

INTERVENTIONS:
Biological: Evolocumab — Administered by subcutaneous injection
  Other Names: AMG 145; Repatha
  Arms: A10 EvoMab Q2W; A10 EvoMab QM; A80 EvoMab Q2W; A80 EvoMab QM; R40 EvoMab Q2W; R40 EvoMab QM; R5 EvoMab Q2W; R5 EvoMab QM; S40 EvoMab Q2W; S40 EvoMab QM
Drug: Ezetimibe — Administered orally once a day
  Other Names: Zetia
  Arms: A10 EZE (Q2W); A10 EZE (QM); A80 EZE (Q2W); A80 EZE (QM)
Drug: Placebo to Evolocumab — Administered by subcutaneous injection
  Arms: A10 EZE (Q2W); A10 EZE (QM); A10 PBO Q2W; A10 PBO QM; A80 EZE (Q2W); A80 EZE (QM); A80 PBO Q2W; A80 PBO QM; R40 PBO Q2W; R40 PBO QM; R5 PBO Q2W; R5 PBO QM; S40 PBO Q2W; S40 PBO QM
Drug: Placebo to Ezetimibe — Administered orally once a day
  Arms: A10 EvoMab Q2W; A10 EvoMab QM; A10 PBO Q2W; A10 PBO QM; A80 EvoMab Q2W; A80 EvoMab QM; A80 PBO Q2W; A80 PBO QM
Drug: Atorvastatin — Administered orally once a day
  Other Names: Lipitor
  Arms: A10 EZE (Q2W); A10 EZE (QM); A10 EvoMab Q2W; A10 EvoMab QM; A10 PBO Q2W; A10 PBO QM; A80 EZE (Q2W); A80 EZE (QM); A80 EvoMab Q2W; A80 EvoMab QM; A80 PBO Q2W; A80 PBO QM
Drug: Rosuvastatin — Administered orally once a day
  Other Names: Crestor
  Arms: R40 EvoMab Q2W; R40 EvoMab QM; R40 PBO Q2W; R40 PBO QM; R5 EvoMab Q2W; R5 EvoMab QM; R5 PBO Q2W; R5 PBO QM
Drug: Simvastatin — Administered orally once a day
  Other Names: Zocor
  Arms: S40 EvoMab Q2W; S40 EvoMab QM; S40 PBO Q2W; S40 PBO QM

SUMMARY:
The primary objective was to evaluate the effect of 12 weeks of evolocumab administered subcutaneously every 2 weeks (Q2W) and monthly (QM) when used in combination with a statin, compared with placebo, on percent change from baseline in low-density lipoprotein cholesterol (LDL-C) in patients with primary hypercholesterolemia and mixed dyslipidemia.

DETAILED DESCRIPTION:
Prior to the first randomization, participants entered a screening period to determine eligibility. During screening, all participants received subcutaneous placebo corresponding to the once monthly dose volume. Participants who completed the screening period and met eligibility criteria were randomized to 1 of 5 open-label statin cohorts (atorvastatin 10 mg or 80 mg, rosuvastatin 5 mg or 40 mg, or simvastatin 40 mg) for a 4 week lipid stabilization period based on statin therapy at the time of study entry (no statin use vs non-intensive statin use vs intensive statin use).

After the 4-week lipid-stabilization period, eligible patients taking rosuvastatin or simvastatin during the lipid-stabilization phase were then randomized to 1 of 4 treatment groups: evolocumab (140 mg, subcutaneous, every 2 weeks) or matching placebo (subcutaneous, every 2 weeks), or evolocumab (420 mg, subcutaneous, monthly) or matching placebo (subcutaneous, monthly). Patients taking atorvastatin during the lipid-stabilization phase were then randomized to 1 of 6 treatment groups: evolocumab (140 mg, subcutaneous, every 2 weeks) and placebo (oral, daily), evolocumab (420 mg, subcutaneous, monthly) and placebo (oral, daily), placebo (subcutaneous, every 2 weeks) and placebo (oral, daily) or ezetimibe (10 mg, oral, daily), or placebo (subcutaneous, monthly) and placebo (oral, daily) or ezetimibe (10 mg, oral, daily).

A participant was considered randomized into the study after successfully completing the screening period, meeting all inclusion/exclusion criteria, and undergoing both randomization procedures.

Participants randomized to simvastatin who were taking verapamil or diltiazem prior to randomization received simvastatin 10 mg once daily (QD) while participants who were taking amlodipine, amiodarone or ranolazine prior to randomization received simvastatin 20 mg QD. All other participants randomized to simvastatin received simvastatin 40 mg QD.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 to ≤ 80 years of age
* Subjects not taking a statin must have fasting LDL-C of at least 150 mg/dL (4.0 mmol/L)
* Subjects already on a non-intensive statin must have fasting LDL-C at screening ≥ 100 mg/dL (2.6 mmol/L)
* Subjects already on a intensive statin must have fasting LDL-C at screening ≥ 80 mg/dL (2.1 mmol/L)
* Fasting triglycerides ≤ 400 mg/dL (4.5 mmol/L)

Exclusion Criteria:

* Statin intolerance
* New York Heart association (NYHA) III or IV heart failure
* Uncontrolled hypertension
* Uncontrolled cardiac arrhythmia
* Type 1 diabetes, poorly controlled type 2 diabetes
* Uncontrolled hypothyroidism or hyperthyroidism

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2067 (Actual)
Dates: Start 2013-01-15 (Actual); Primary Completion 2013-11-12 (Actual); Study Completion 2013-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (214):
- United States (61):
  - Research Site, Birmingham, Alabama
  - Research Site, Glendale, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Carmichael, California
  - Research Site, Encino, California
  - Research Site, Long Beach, California
  - Research Site, Newport Beach, California
  - Research Site, San Diego, California
  - Research Site, Santa Ana, California
  - Research Site, Santa Rosa, California
  - Research Site, Thousand Oaks, California
  - Research Site, Torrance, California
  - Research Site, Tustin, California
  - Research Site, Westlake Village, California
  - Research Site, Littleton, Colorado
  - Research Site, Daytona Beach, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Melbourne, Florida
  - Research Site, Miami, Florida
  - Research Site, Port Charlotte, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Boise, Idaho
  - Research Site, Hammond, Indiana
  - Research Site, Indianapolis, Indiana
  - Research Site, Valparaiso, Indiana
  - Research Site, Iowa City, Iowa
  - Research Site, Crestview Hills, Kentucky
  - Research Site, Monroe, Louisiana
  - Research Site, Auburn, Maine
  - Research Site, Bangor, Maine
  - Research Site, Portland, Maine
  - Research Site, Baltimore, Maryland
  - Research Site, Ypsilanti, Michigan
  - Research Site, Tupelo, Mississippi
  - Research Site, Billings, Montana
  - Research Site, Voorhees Township, New Jersey
  - Research Site, Manlius, New York
  - Research Site, Rochester, New York
  - Research Site, Syracuse, New York
  - Research Site, Williamsville, New York
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cadiz, Ohio
  - Research Site, Canton, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Mansfield, Ohio
  - Research Site, Marion, Ohio
  - Research Site, Sandusky, Ohio
  - Research Site, Norman, Oklahoma
  - Research Site, Duncansville, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, York, Pennsylvania
  - Research Site, Florence, South Carolina
  - Research Site, Rapid City, South Dakota
  - Research Site, Jackson, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Suffolk, Virginia
  - Research Site, Winchester, Virginia
  - Research Site, Tacoma, Washington
- Australia (6):
  - Research Site, Sydney, New South Wales
  - Research Site, Ashford, South Australia
  - Research Site, Fullarton, South Australia
  - Research Site, Fitzroy, Victoria
  - Research Site, Heidelberg Heights, Victoria
  - Research Site, Richmond, Victoria
- Belgium (6):
  - Research Site, Blankenberge
  - Research Site, ChÃªnÃ©e
  - Research Site, Hasselt
  - Research Site, Ostend
  - Research Site, Tremelo
  - Research Site, Vilvoorde
- Canada (19):
  - Research Site, Burnaby, British Columbia
  - Research Site, Kelowna, British Columbia
  - Research Site, Surrey, British Columbia
  - Research Site, Saint Johnâ€™s, Newfoundland and Labrador
  - Research Site, Cambridge, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, London, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, Oshawa, Ontario
  - Research Site, Sarnia, Ontario
  - Research Site, Scarborough Village, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Woodstock, Ontario
  - Research Site, Brossard, Quebec
  - Research Site, Greenfield Park, Quebec
  - Research Site, Lachine, Quebec
  - Research Site, Longueuil, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Pointe-Claire, Quebec
- Czechia (10):
  - Research Site, Brno
  - Research Site, Kladno
  - Research Site, Litoměřice
  - Research Site, Moravské Budějovice
  - Research Site, Olomouc
  - Research Site, Pardubice
  - Research Site, Prague
  - Research Site, Slaný
  - Research Site, Svitavy
  - Research Site, Ústí nad Orlicí
- Denmark (3):
  - Research Site, Aalborg
  - Research Site, Ballerup Municipality
  - Research Site, Vejle
- France (9):
  - Research Site, Brest
  - Research Site, Caen
  - Research Site, Dijon
  - Research Site, Le Creusot
  - Research Site, Montpellier
  - Research Site, Nantes
  - Research Site, Paris
  - Research Site, Poitiers
  - Research Site, Strasbourg
- Germany (10):
  - Research Site, Bad Krozingen
  - Research Site, Berlin
  - Research Site, Freiburg im Breisgau
  - Research Site, Heidelberg
  - Research Site, Hellersdorf
  - Research Site, Homburg
  - Research Site, Leipzig
  - Research Site, Magdeburg
  - Research Site, Messkirch
  - Research Site, Witten
- Hong Kong (2):
  - Research Site, Hong Kong
  - Research Site, New Territories
- Hungary (11):
  - Research Site, Baja
  - Research Site, Berettyóújfalu
  - Research Site, Dunaújváros
  - Research Site, Eger
  - Research Site, Gyöngyös
  - Research Site, Hódmezővásárhely
  - Research Site, Jászberény
  - Research Site, Komárom
  - Research Site, Marcali
  - Research Site, Mosonmagyaróvár
  - Research Site, Pécs
- Italy (10):
  - Research Site, Bologna
  - Research Site, Cagliari
  - Research Site, Chieti
  - Research Site, Ferrara
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Padua
  - Research Site, Perugia
  - Research Site, Pisa
  - Research Site, Trieste
- Mexico (7):
  - Research Site, León, Guanajuato
  - Research Site, Guadalajara, Jalisco
  - Research Site, Mexico City, Mexico City
  - Research Site, Monterrey, Nuevo LeÃ³n
  - Research Site, San Luis Potosí City, San Luis PotosÃ-
  - Research Site, Tampico, Tamaulipas
  - Research Site, Durango
- Netherlands (9):
  - Research Site, Amsterdam
  - Research Site, Den Helder
  - Research Site, Groningen
  - Research Site, Hoogeveen
  - Research Site, Nieuwegein
  - Research Site, Nijmegen
  - Research Site, Rotterdam
  - Research Site, Waalwijk
  - Research Site, Zwijndrecht
- Russia (6):
  - Research Site, Barnaul
  - Research Site, Kemerovo
  - Research Site, Moscow
  - Research Site, Novosibirsk
  - Research Site, Saint Petersburg
  - Research Site, Saratov
- South Africa (8):
  - Research Site, Alberton, Gauteng
  - Research Site, Johannesburg, Gauteng
  - Research Site, Lyttelton, Gauteng
  - Research Site, Pretoria, Gauteng
  - Research Site, Kuils River, Western Cape
  - Research Site, Somerset West, Western Cape
  - Research Site, Bloemfontein
  - Research Site, Cape Town
- South Korea (2):
  - Research Site, Seoul
  - Research Site, Suwon
- Spain (8):
  - Research Site, AlmerÃ-a, AndalucÃ-a
  - Research Site, Almería, AndalucÃ-a
  - Research Site, Barcelona, CataluÃ±a
  - Research Site, L'Hospitalet de Llobregat, CataluÃ±a
  - Research Site, Pozuelo de AlarcÃ³n, Madrid
  - Research Site, Pozuelo de Alarcón, Madrid
  - Research Site, Valencia, Valencia
  - Research Site, Madrid
- Sweden (5):
  - Research Site, Ã-rebro
  - Research Site, GÃ¶teborg
  - Research Site, Lund
  - Research Site, Stockholm
  - Research Site, Uddevalla
- Switzerland (6):
  - Research Site, Bellinzona
  - Research Site, Geneva
  - Research Site, Lausanne
  - Research Site, Muensterlingen
  - Research Site, Sankt Gallen
  - Research Site, Zurich
- Taiwan (2):
  - Research Site, Kaohsiung City
  - Research Site, Taipei
- United Kingdom (14):
  - Research Site, Birmingham
  - Research Site, Blackpool
  - Research Site, Cardiff
  - Research Site, Chesterfield
  - Research Site, Chorley
  - Research Site, Doncaster
  - Research Site, Glasgow
  - Research Site, Harrow
  - Research Site, Liverpool
  - Research Site, Manchester
  - Research Site, Reading
  - Research Site, Scunthorpe
  - Research Site, Wakefield
  - Research Site, Whitby

REFERENCES:
- [Background] Robinson JG, Nedergaard BS, Rogers WJ, Fialkow J, Neutel JM, Ramstad D, Somaratne R, Legg JC, Nelson P, Scott R, Wasserman SM, Weiss R; LAPLACE-2 Investigators. Effect of evolocumab or ezetimibe added to moderate- or high-intensity statin therapy on LDL-C lowering in patients with hypercholesterolemia: the LAPLACE-2 randomized clinical trial. JAMA. 2014 May 14;311(18):1870-82. doi: 10.1001/jama.2014.4030. PMID 24825642
- [Background] Robinson JG, Rogers WJ, Nedergaard BS, Fialkow J, Neutel JM, Ramstad D, Somaratne R, Legg JC, Nelson P, Scott R, Wasserman SM, Weiss R. Rationale and design of LAPLACE-2: a phase 3, randomized, double-blind, placebo- and ezetimibe-controlled trial evaluating the efficacy and safety of evolocumab in subjects with hypercholesterolemia on background statin therapy. Clin Cardiol. 2014 Apr;37(4):195-203. doi: 10.1002/clc.22252. Epub 2014 Jan 30. PMID 24481874
- [Background] Daviglus ML, Ferdinand KC, Lopez JAG, Wu Y, Monsalvo ML, Rodriguez CJ. Effects of Evolocumab on Low-Density Lipoprotein Cholesterol, Non-High Density Lipoprotein Cholesterol, Apolipoprotein B, and Lipoprotein(a) by Race and Ethnicity: A Meta-Analysis of Individual Participant Data From Double-Blind and Open-Label Extension Studies. J Am Heart Assoc. 2021 Jan 5;10(1):e016839. doi: 10.1161/JAHA.120.016839. Epub 2020 Dec 16. PMID 33325247
- [Background] Koren MJ, Jones PH, Robinson JG, Sullivan D, Cho L, Hucko T, Lopez JAG, Fleishman AN, Somaratne R, Stroes E. A Comparison of Ezetimibe and Evolocumab for Atherogenic Lipid Reduction in Four Patient Populations: A Pooled Efficacy and Safety Analysis of Three Phase 3 Studies. Cardiol Ther. 2020 Dec;9(2):447-465. doi: 10.1007/s40119-020-00181-8. Epub 2020 Jun 20. PMID 32564340
- [Background] Kuchimanchi M, Grover A, Emery MG, Somaratne R, Wasserman SM, Gibbs JP, Doshi S. Population pharmacokinetics and exposure-response modeling and simulation for evolocumab in healthy volunteers and patients with hypercholesterolemia. J Pharmacokinet Pharmacodyn. 2018 Jun;45(3):505-522. doi: 10.1007/s10928-018-9592-y. Epub 2018 May 7. PMID 29736889
- [Background] Kasichayanula S, Grover A, Emery MG, Gibbs MA, Somaratne R, Wasserman SM, Gibbs JP. Clinical Pharmacokinetics and Pharmacodynamics of Evolocumab, a PCSK9 Inhibitor. Clin Pharmacokinet. 2018 Jul;57(7):769-779. doi: 10.1007/s40262-017-0620-7. PMID 29353350
- [Background] Shapiro MD, Minnier J, Tavori H, Kassahun H, Flower A, Somaratne R, Fazio S. Relationship Between Low-Density Lipoprotein Cholesterol and Lipoprotein(a) Lowering in Response to PCSK9 Inhibition With Evolocumab. J Am Heart Assoc. 2019 Feb 19;8(4):e010932. doi: 10.1161/JAHA.118.010932. PMID 30755061
- [Background] Stroes E, Robinson JG, Raal FJ, Dufour R, Sullivan D, Kassahun H, Ma Y, Wasserman SM, Koren MJ. Consistent LDL-C response with evolocumab among patient subgroups in PROFICIO: A pooled analysis of 3146 patients from phase 3 studies. Clin Cardiol. 2018 Oct;41(10):1328-1335. doi: 10.1002/clc.23049. Epub 2018 Oct 21. PMID 30120772
- [Background] Toth PP, Descamps O, Genest J, Sattar N, Preiss D, Dent R, Djedjos C, Wu Y, Geller M, Uhart M, Somaratne R, Wasserman SM; PROFICIO Investigators. Pooled Safety Analysis of Evolocumab in Over 6000 Patients From Double-Blind and Open-Label Extension Studies. Circulation. 2017 May 9;135(19):1819-1831. doi: 10.1161/CIRCULATIONAHA.116.025233. Epub 2017 Mar 1. PMID 28249876
- [Background] Toth PP, Jones SR, Monsalvo ML, Elliott-Davey M, Lopez JAG, Banach M. Effect of Evolocumab on Non-High-Density Lipoprotein Cholesterol, Apolipoprotein B, and Lipoprotein(a): A Pooled Analysis of Phase 2 and Phase 3 Studies. J Am Heart Assoc. 2020 Mar 3;9(5):e014129. doi: 10.1161/JAHA.119.014129. Epub 2020 Mar 2. PMID 32114889
- [Background] Wasserman SM, Sabatine MS, Koren MJ, Giugliano RP, Legg JC, Emery MG, Doshi S, Liu T, Somaratne R, Gibbs JP. Comparison of LDL-C Reduction Using Different Evolocumab Doses and Intervals: Biological Insights and Treatment Implications. J Cardiovasc Pharmacol Ther. 2018 Sep;23(5):423-432. doi: 10.1177/1074248418774043. Epub 2018 May 16. PMID 29768954
- [Background] May HT, Muhlestein JB, Ma Y, Lopez JAG, Coll B, Nelson J. Effects of Evolocumab on the ApoA1 Remnant Ratio: A Pooled Analysis of Phase 3 Studies. Cardiol Ther. 2019 Jun;8(1):91-102. doi: 10.1007/s40119-019-0133-6. Epub 2019 Mar 9. PMID 30852766
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adults aged 18 to 80 years with screening low-density lipoprotein cholesterol (LDL-C) ≥ 150 mg/dL (no statin at screening), ≥ 100 mg/dL (non-intensive statin at screening), or ≥ 80 mg/dL (intensive statin at screening) and fasting triglycerides ≤ 400 mg/dL.
  First patient enrolled on 15 January 2013; Last patient enrolled on 10 July 2013.
Pre-assignment Details: 2067 patients were first randomized to 1 of the 5 open-label statin cohorts (atorvastatin 10 mg or 80 mg, rosuvastatin 5 mg or 40 mg, or simvastatin 40 mg); 1899 were then randomized to blinded investigational product.
  Randomization into the statin dose cohorts was stratified by entry statin therapy and by use of certain concomitant medications.
Groups:
- A10 PBO QM: Participants received atorvastatin 10 mg a day during the 4-week lipid stabilization period and then in combination with placebo subcutaneous injection once a month (QM) and placebo tablets once daily for up to 12 weeks.
- A10 EZE (Q2W): Participants received atorvastatin 10 mg a day during the 4-week lipid stabilization period and then in combination with placebo subcutaneous injection once every 2 weeks and 10 mg ezetimibe (EZE) orally once daily for up to 12 weeks.
- A10 EZE (QM): Participants received atorvastatin 10 mg a day during the 4-week lipid stabilization period and then in combination with placebo subcutaneous injection once a month and 10 mg ezetimibe orally once daily for up to 12 weeks.
- A10 EvoMab Q2W: Participants received atorvastatin 10 mg a day during the 4-week lipid stabilization period and then in combination with 140 mg evolocumab (EvoMab) by subcutaneous injection once every 2 weeks and placebo tablets once daily for up to 12 weeks.
- A10 EvoMab QM: Participants received atorvastatin 10 mg a day during the 4-week lipid stabilization period and then in combination with 420 mg evolocumab by subcutaneous injection once a month and placebo tablets once daily for up to 12 weeks.
- A80 PBO Q2W: Participants received atorvastatin 80 mg a day during the 4-week lipid stabilization period and then in combination with placebo subcutaneous injection once every 2 weeks and placebo tablets once daily for up to 12 weeks.
- A80 PBO QM: Participants received atorvastatin 80 mg a day during the 4-week lipid stabilization period and then in combination with placebo subcutaneous injection once a month and placebo tablets once daily for up to 12 weeks.
- A80 EZE (Q2W): Participants received atorvastatin 80 mg a day during the 4-week lipid stabilization period and then in combination with placebo subcutaneous injection once every 2 weeks and 10 mg ezetimibe orally once daily for up to 12 weeks.
- A80 EZE (QM): Participants received atorvastatin 80 mg a day during the 4-week lipid stabilization period and then in combination with placebo subcutaneous injection once a month and 10 mg ezetimibe orally once daily for up to 12 weeks.
- A80 EvoMab Q2W: Participants received atorvastatin 80 mg a day during the 4-week lipid stabilization period and then in combination with 140 mg evolocumab by subcutaneous injection once every 2 weeks and placebo tablets once daily for up to 12 weeks.
- A80 EvoMab QM: Participants received atorvastatin 80 mg a day during the 4-week lipid stabilization period and then in combination with 420 mg evolocumab by subcutaneous injection once a month and placebo tablets once daily for up to 12 weeks.
- R5 PBO Q2W: Participants received rosuvastatin 5 mg a day during the 4-week lipid stabilization period and then in combination with placebo subcutaneous injection once every 2 weeks for up to 12 weeks.
- R5 PBO QM: Participants received rosuvastatin 5 mg a day during the 4-week lipid stabilization period and then in combination with placebo subcutaneous injection once a month for up to 12 weeks.
- R5 EvoMab Q2W: Participants received rosuvastatin 5 mg a day during the 4-week lipid stabilization period and then in combination with 140 mg evolocumab by subcutaneous injection once every 2 weeks for up to 12 weeks.
- R5 EvoMab QM: Participants received rosuvastatin 5 mg a day during the 4-week lipid stabilization period and then in combination with 420 mg evolocumab by subcutaneous injection once a month for up to 12 weeks.
- R40 PBO Q2W: Participants received rosuvastatin 40 mg a day during the 4-week lipid stabilization period and then in combination with placebo subcutaneous injection once every 2 weeks for up to 12 weeks.
- R40 PBO QM: Participants received rosuvastatin 40 mg a day during the 4-week lipid stabilization period and then in combination with placebo subcutaneous injection once a month for up to 12 weeks.
- R40 EvoMab Q2W: Participants received rosuvastatin 40 mg a day during the 4-week lipid stabilization period and then in combination with 140 mg evolocumab by subcutaneous injection once every 2 weeks for up to 12 weeks.
- R40 EvoMab QM: Participants received rosuvastatin 40 mg a day during the 4-week lipid stabilization period and then in combination with 420 mg evolocumab by subcutaneous injection once a month for up to 12 weeks.
- S40 PBO Q2W: Participants received simvastatin 40 mg a day during the 4-week lipid stabilization period and then in combination with placebo subcutaneous injection once every 2 weeks for up to 12 weeks.
- S40 PBO QM: Participants received simvastatin 40 mg a day during the 4-week lipid stabilization period and then in combination with placebo subcutaneous injection once a month for up to 12 weeks.
- S40 EvoMab Q2W: Participants received simvastatin 40 mg a day during the 4-week lipid stabilization period and then in combination with 140 mg evolocumab by subcutaneous injection once every 2 weeks for up to 12 weeks.
- S40 EvoMab QM: Participants received simvastatin 40 mg a day during the 4-week lipid stabilization period and then in combination with 420 mg evolocumab by subcutaneous injection once a month for up to 12 weeks.
Period: Overall Study
Arm/Group | A10 PBO Q2W | A10 PBO QM | A10 EZE (Q2W) | A10 EZE (QM) | A10 EvoMab Q2W | A10 EvoMab QM | A80 PBO Q2W | A80 PBO QM | A80 EZE (Q2W) | A80 EZE (QM) | A80 EvoMab Q2W | A80 EvoMab QM | R5 PBO Q2W | R5 PBO QM | R5 EvoMab Q2W | R5 EvoMab QM | R40 PBO Q2W | R40 PBO QM | R40 EvoMab Q2W | R40 EvoMab QM | S40 PBO Q2W | S40 PBO QM | S40 EvoMab Q2W | S40 EvoMab QM
Started | 56 | 55 | 56 | 55 | 110 | 110 | 55 | 55 | 56 | 54 | 110 | 110 | 58 | 57 | 114 | 115 | 56 | 56 | 111 | 112 | 56 | 55 | 112 | 115
Received Treatment | 56 | 55 | 56 | 55 | 110 | 110 | 55 | 55 | 56 | 54 | 109 | 110 | 58 | 57 | 113 | 115 | 56 | 55 | 111 | 112 | 56 | 55 | 112 | 115
Completed | 54 | 54 | 51 | 55 | 108 | 107 | 48 | 55 | 53 | 53 | 102 | 108 | 54 | 57 | 102 | 112 | 55 | 55 | 105 | 110 | 52 | 54 | 109 | 113
Not Completed | 2 | 1 | 5 | 0 | 2 | 3 | 7 | 0 | 3 | 1 | 8 | 2 | 4 | 0 | 12 | 3 | 1 | 1 | 6 | 2 | 4 | 1 | 3 | 2
Not completed — Withdrawal by Subject | 2 | 1 | 4 | 0 | 0 | 3 | 4 | 0 | 1 | 1 | 2 | 2 | 2 | 0 | 6 | 3 | 0 | 1 | 1 | 1 | 2 | 1 | 2 | 1
Not completed — Decision by sponsor | 0 | 0 | 1 | 0 | 2 | 0 | 2 | 0 | 2 | 0 | 6 | 0 | 1 | 0 | 5 | 0 | 0 | 0 | 4 | 0 | 2 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A10 PBO Q2W | A10 PBO QM | A10 EZE (Q2W) | A10 EZE (QM) | A10 EvoMab Q2W | A10 EvoMab QM | A80 PBO Q2W | A80 PBO QM | A80 EZE (Q2W) | A80 EZE (QM) | A80 EvoMab Q2W | A80 EvoMab QM | R5 PBO Q2W | R5 PBO QM | R5 EvoMab Q2W | R5 EvoMab QM | R40 PBO Q2W | R40 PBO QM | R40 EvoMab Q2W | R40 EvoMab QM | S40 PBO Q2W | S40 PBO QM | S40 EvoMab Q2W | S40 EvoMab QM | Total
Number analyzed (Participants) | 56 | 55 | 56 | 55 | 110 | 110 | 55 | 55 | 56 | 54 | 110 | 110 | 58 | 57 | 114 | 115 | 56 | 56 | 111 | 112 | 56 | 55 | 112 | 115 | 1899
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (10.5) | 62.2 (10.4) | 61.0 (9.0) | 60.6 (9.2) | 58.3 (8.4) | 59.6 (11.1) | 57.1 (9.9) | 58.8 (11.5) | 60.5 (10.2) | 61.1 (8.9) | 59.7 (10.2) | 60.1 (10.2) | 61.2 (9.1) | 59.6 (9.2) | 58.9 (11.2) | 59.3 (10.5) | 60.2 (8.7) | 58.3 (11.3) | 59.5 (9.2) | 59.6 (9.0) | 61.9 (9.7) | 61.5 (10.3) | 59.7 (9.2) | 61.5 (9.6) | 59.8 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 28 | 29 | 28 | 56 | 44 | 22 | 24 | 24 | 28 | 44 | 48 | 35 | 27 | 52 | 51 | 21 | 27 | 43 | 52 | 32 | 28 | 45 | 59 | 871
  Male | 32 | 27 | 27 | 27 | 54 | 66 | 33 | 31 | 32 | 26 | 66 | 62 | 23 | 30 | 62 | 64 | 35 | 29 | 68 | 60 | 24 | 27 | 67 | 56 | 1028
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 3 | 2 | 2 | 1 | 5 | 2 | 5 | 5 | 4 | 4 | 5 | 7 | 2 | 4 | 6 | 3 | 2 | 3 | 6 | 5 | 1 | 2 | 3 | 5 | 87
  Not Hispanic or Latino | 53 | 53 | 54 | 54 | 105 | 108 | 50 | 50 | 52 | 50 | 105 | 103 | 56 | 53 | 108 | 112 | 54 | 53 | 105 | 107 | 55 | 53 | 109 | 110 | 1812
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Asian | 1 | 0 | 2 | 1 | 3 | 4 | 1 | 0 | 0 | 3 | 1 | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 25
  Black or African American | 3 | 0 | 1 | 2 | 9 | 4 | 1 | 2 | 3 | 4 | 3 | 4 | 2 | 1 | 7 | 5 | 0 | 3 | 5 | 3 | 3 | 1 | 4 | 5 | 75
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 4
  White | 52 | 55 | 53 | 52 | 97 | 101 | 51 | 52 | 53 | 46 | 105 | 105 | 56 | 56 | 104 | 107 | 55 | 52 | 105 | 109 | 49 | 54 | 106 | 110 | 1785
  Other | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 7
  Mixed Race | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Stratification Factor: Entry Statin Therapy [Number; unit: participants] — Intensive statin use was defined as daily atorvastatin (40 mg or greater), rosuvastatin (20 mg or greater), simvastatin (80 mg), or any statin plus ezetimibe.
  participants
    Intensive statin use | 18 | 19 | 10 | 14 | 28 | 35 | 15 | 12 | 21 | 11 | 34 | 35 | 13 | 13 | 33 | 38 | 13 | 13 | 33 | 37 | 19 | 13 | 31 | 34 | 542
    Non-intensive statin use | 20 | 25 | 30 | 21 | 52 | 40 | 22 | 27 | 22 | 21 | 47 | 46 | 25 | 28 | 49 | 42 | 23 | 22 | 50 | 44 | 21 | 26 | 45 | 48 | 796
    No statin use | 18 | 11 | 16 | 20 | 30 | 35 | 18 | 16 | 13 | 22 | 29 | 29 | 20 | 16 | 32 | 35 | 20 | 21 | 28 | 31 | 16 | 16 | 36 | 33 | 561
Low-Density Lipoprotein Cholesterol (LDL-C) Concentration [Mean (Standard Deviation); unit: mg/dL] — Data are provided for the full analysis set (all participants randomized to investigational product (IP) who received at least 1 dose of IP (subcutaneously or orally). Baseline was measured after the lipid stabilization period and before administration of first dose of study drug.
  mg/dL | 123.0 (46.6) | 123.7 (47.9) | 126.8 (49.6) | 119.3 (28.1) | 124.2 (43.4) | 126.1 (50.4) | 100.3 (36.2) | 94.7 (31.9) | 98.7 (34.0) | 92.3 (19.3) | 94.2 (34.8) | 93.8 (32.3) | 115.6 (39.8) | 119.9 (39.1) | 118.7 (40.9) | 122.9 (42.0) | 77.4 (20.9) | 102.9 (49.3) | 88.5 (31.5) | 88.5 (31.3) | 110.3 (28.0) | 108.6 (30.9) | 114.9 (34.5) | 123.7 (48.5) | 109.1 (41.1)
Non-High-Density Lipoprotein Cholesterol (non-HDL-C) Concentration [Mean (Standard Deviation); unit: mg/dL] — Data are provided for the full analysis set. Baseline was measured after the lipid stabilization period and before administration of first dose of study drug.
  mg/dL | 149.1 (46.9) | 147.7 (51.4) | 153.8 (53.2) | 148.3 (36.8) | 152.3 (45.6) | 154.3 (53.1) | 124.2 (39.3) | 116.5 (35.7) | 124.8 (35.4) | 118.4 (25.5) | 120.2 (42.3) | 117.2 (36.3) | 141.1 (41.6) | 148.3 (43.3) | 146.6 (43.2) | 152.0 (46.4) | 103.9 (25.7) | 128.7 (53.4) | 113.5 (36.0) | 114.3 (34.7) | 138.4 (29.3) | 135.7 (38.4) | 146.8 (41.8) | 151.2 (51.5) | 150.3 (27.6)
Apolipoprotein B Concentration [Mean (Standard Deviation); unit: mg/dL] — Data are provided for the full analysis set. Baseline was measured after the lipid stabilization period and before administration of first dose of study drug.
  mg/dL | 95.3 (26.0) | 95.3 (29.6) | 101.3 (31.2) | 94.6 (20.4) | 99.7 (26.4) | 97.3 (28.9) | 81.1 (22.1) | 80.1 (21.4) | 85.3 (23.1) | 78.7 (16.9) | 79.9 (25.1) | 77.9 (21.5) | 93.1 (27.3) | 95.9 (25.2) | 95.4 (27.0) | 97.2 (26.9) | 71.0 (16.6) | 84.8 (29.7) | 77.4 (22.3) | 78.7 (23.1) | 91.6 (18.4) | 89.8 (20.7) | 94.2 (24.0) | 96.5 (27.5) | 89.1 (26.1)
Total Cholesterol/HDL-C Ratio [Mean (Standard Deviation); unit: ratio] — Data are provided for the full analysis set. Baseline was measured after the lipid stabilization period and before administration of first dose of study drug.
  ratio | 3.988 (1.154) | 3.859 (1.396) | 4.112 (1.311) | 4.002 (1.100) | 3.980 (1.224) | 4.100 (1.636) | 3.704 (1.260) | 3.461 (1.093) | 3.748 (1.099) | 3.540 (1.100) | 3.696 (1.371) | 3.462 (1.000) | 4.044 (1.685) | 3.891 (1.234) | 3.915 (1.216) | 4.178 (1.932) | 3.086 (0.728) | 3.547 (1.355) | 3.413 (1.355) | 3.307 (1.061) | 3.733 (1.079) | 3.595 (1.345) | 4.196 (1.436) | 3.924 (1.420) | 3.786 (1.353)
Apolipoprotein B/Apolipoprotein A1 Ratio [Mean (Standard Deviation); unit: ratio] — Data are provided for the full analysis set. Baseline was measured after the lipid stabilization period and before administration of first dose of study drug.
  ratio | 0.666 (0.216) | 0.647 (0.266) | 0.692 (0.243) | 0.640 (0.169) | 0.663 (0.217) | 0.659 (0.249) | 0.603 (0.221) | 0.571 (0.189) | 0.640 (0.234) | 0.560 (0.157) | 0.593 (0.227) | 0.562 (0.171) | 0.661 (0.273) | 0.636 (0.207) | 0.640 (0.249) | 0.676 (0.341) | 0.479 (0.129) | 0.562 (0.217) | 0.538 (0.227) | 0.536 (0.193) | 0.611 (0.179) | 0.581 (0.174) | 0.657 (0.193) | 0.639 (0.224) | 0.614 (0.229)
Lipoprotein(a) Concentration [Median (Inter-Quartile Range); unit: nmol/L] — Data are provided for the full analysis set. Baseline was measured after the lipid stabilization period and before administration of first dose of study drug.
  nmol/L | 31.5 [13.0 to 87.5] | 41.0 [15.0 to 106.0] | 37.0 [9.5 to 190.0] | 33.0 [8.0 to 163.0] | 27.0 [8.0 to 120.0] | 49.0 [11.0 to 169.0] | 53.0 [15.0 to 177.0] | 50.0 [13.0 to 152.0] | 25.0 [12.0 to 108.0] | 61.5 [12.0 to 192.0] | 32.0 [11.5 to 135.5] | 24.5 [8.0 to 93.0] | 34.0 [8.0 to 158.0] | 35.0 [14.0 to 156.5] | 38.0 [11.0 to 165.0] | 32.0 [9.0 to 172.0] | 28.5 [7.0 to 171.0] | 33.0 [11.0 to 148.0] | 41.0 [10.0 to 183.0] | 49.5 [11.0 to 184.5] | 36.5 [17.5 to 140.5] | 28.0 [13.0 to 180.0] | 32.5 [13.0 to 157.0] | 37.0 [11.0 to 141.0] | 34.0 [11.0 to 161.5]
Triglyceride Concentration [Median (Inter-Quartile Range); unit: mg/dL] — Data are provided for the full analysis set. Baseline was measured after the lipid stabilization period and before administration of first dose of study drug.
  mg/dL | 112.0 [83.0 to 176.0] | 108.0 [83.0 to 145.0] | 129.5 [94.0 to 151.5] | 119.0 [87.0 to 168.0] | 135.0 [99.0 to 189.0] | 119.0 [84.0 to 161.0] | 104.0 [82.0 to 142.0] | 104.0 [76.0 to 124.0] | 133.0 [89.0 to 155.0] | 109.0 [80.0 to 171.0] | 104.0 [81.0 to 163.0] | 106.5 [79.0 to 137.0] | 112.5 [89.0 to 148.0] | 134.0 [86.0 to 184.0] | 116.0 [90.0 to 168.0] | 121.0 [93.0 to 161.0] | 128.0 [91.5 to 162.0] | 116.0 [78.0 to 160.0] | 102.0 [79.0 to 151.0] | 119.5 [87.0 to 149.5] | 124.0 [90.0 to 173.0] | 106.0 [87.0 to 139.0] | 129.0 [91.5 to 195.0] | 110.0 [84.0 to 161.0] | 116.0 [86.0 to 158.0]
Very Low Density Lipoprotein Cholesterol (VLDL-C) Concentration [Median (Inter-Quartile Range); unit: mg/dL] — Data are provided for the full analysis set. Baseline was measured after the lipid stabilization period and before administration of first dose of study drug.
  mg/dL | 22.0 [17.0 to 35.0] | 22.0 [17.0 to 29.0] | 25.5 [19.0 to 30.0] | 24.0 [17.0 to 33.0] | 27.0 [20.0 to 38.0] | 24.0 [17.0 to 32.0] | 21.0 [16.0 to 28.0] | 21.0 [15.0 to 25.0] | 26.5 [18.0 to 31.0] | 22.0 [16.0 to 34.0] | 21.0 [16.0 to 33.0] | 21.0 [16.0 to 27.0] | 22.5 [18.0 to 30.0] | 27.0 [17.0 to 37.0] | 23.0 [18.0 to 34.0] | 24.0 [19.0 to 32.0] | 26.0 [18.5 to 32.5] | 23.0 [16.0 to 32.0] | 20.0 [16.0 to 30.0] | 24.0 [17.0 to 30.0] | 25.0 [18.0 to 34.5] | 21.0 [17.0 to 26.0] | 26.0 [18.5 to 39.0] | 22.0 [17.0 to 32.0] | 23.0 [17.0 to 32.0]
HDL-C Concentration [Mean (Standard Deviation); unit: mg/dL] — Data are provided for the full anlaysis set. Baseline was measured after the lipid stabilization period and before administration of first dose of study drug.
  mg/dL | 54.1 (16.6) | 57.9 (18.4) | 54.1 (17.2) | 52.7 (13.7) | 56.0 (17.9) | 56.1 (17.8) | 50.6 (15.6) | 50.9 (13.0) | 48.7 (12.6) | 51.6 (15.1) | 48.5 (12.9) | 50.8 (13.5) | 52.1 (14.9) | 55.5 (16.0) | 54.5 (15.0) | 54.0 (16.0) | 52.8 (12.9) | 56.0 (18.7) | 53.2 (16.4) | 53.8 (14.6) | 55.0 (14.2) | 59.9 (21.8) | 49.7 (12.6) | 57.3 (17.4) | 53.5 (15.9)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Low-Density Lipoprotein Cholesterol (LDL-C) at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | A10 PBO Q2W | A10 PBO QM | A10 EZE (Q2W) | A10 EZE (QM) | A10 EvoMab Q2W | A10 EvoMab QM | A80 PBO Q2W | A80 PBO QM | A80 EZE (Q2W) | A80 EZE (QM) | A80 EvoMab Q2W | A80 EvoMab QM | R5 PBO Q2W | R5 PBO QM | R5 EvoMab Q2W | R5 EvoMab QM | R40 PBO Q2W | R40 PBO QM | R40 EvoMab Q2W | R40 EvoMab QM | S40 PBO Q2W | S40 PBO QM | S40 EvoMab Q2W | S40 EvoMab QM
Number analyzed (Participants) | 56 | 55 | 56 | 55 | 110 | 110 | 55 | 55 | 56 | 54 | 109 | 110 | 58 | 57 | 113 | 115 | 56 | 55 | 111 | 112 | 56 | 55 | 112 | 115
percent change | 9.86 (2.53) | 0.97 (2.82) | -21.96 (2.63) | -17.08 (2.78) | -61.56 (1.81) | -58.19 (1.99) | 14.49 (4.42) | 11.83 (3.85) | -14.60 (4.29) | -19.80 (3.85) | -61.80 (3.04) | -58.68 (2.74) | 8.12 (2.68) | 5.10 (2.62) | -60.09 (1.94) | -59.40 (1.87) | 9.42 (3.60) | 2.59 (4.30) | -58.89 (2.58) | -52.40 (2.98) | 4.70 (3.61) | 3.40 (4.94) | -65.86 (3.05) | -57.02 (3.93)
Statistical Analysis 1: Comparison: A10 PBO Q2W vs A10 EvoMab Q2W; The null hypothesis was that there was no difference in the percent change from Baseline at Week 12 in LDL-C between evolocumab and placebo, and the alternative hypothesis was that a mean difference did exist; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; The model included treatment group, stratification factors, scheduled visit and the interaction of treatment with scheduled visit; LS Mean Treatment Difference = -71.42, 95% CI 2-sided [-77.55 to -65.29], Standard Error of Mean 3.11
Statistical Analysis 2: Comparison: A10 PBO QM vs A10 EvoMab QM; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -59.16, 95% CI 2-sided [-65.94 to -52.38], Standard Error of Mean 3.44
Statistical Analysis 3: Comparison: A10 EZE (Q2W) vs A10 EvoMab Q2W; The null hypothesis was that there was no mean difference in the percent change from Baseline at Week 12 in LDL-C between evolocumab and ezetimibe, and the alternative hypothesis was that a mean difference did exist; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -39.60, 95% CI 2-sided [-45.81 to -33.40], Standard Error of Mean 3.15
Statistical Analysis 4: Comparison: A10 EZE (QM) vs A10 EvoMab QM; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -41.10, 95% CI 2-sided [-47.83 to -34.37], Standard Error of Mean 3.41
Statistical Analysis 5: Comparison: A80 PBO Q2W vs A80 EvoMab Q2W; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -76.29, 95% CI 2-sided [-86.87 to -65.72], Standard Error of Mean 5.36
Statistical Analysis 6: Comparison: A80 PBO QM vs A80 EvoMab QM; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -70.51, 95% CI 2-sided [-79.81 to -61.20], Standard Error of Mean 4.72
Statistical Analysis 7: Comparison: A80 EZE (Q2W) vs A80 EvoMab Q2W; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -47.20, 95% CI 2-sided [-57.54 to -36.86], Standard Error of Mean 5.24
Statistical Analysis 8: Comparison: A80 EZE (QM) vs A80 EvoMab QM; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -38.88, 95% CI 2-sided [-48.21 to -29.56], Standard Error of Mean 4.73
Statistical Analysis 9: Comparison: R5 PBO Q2W vs R5 EvoMab Q2W; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -68.21, 95% CI 2-sided [-74.72 to -61.70], Standard Error of Mean 3.30
Statistical Analysis 10: Comparison: R5 PBO QM vs R5 EvoMab QM; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -64.49, 95% CI 2-sided [-70.84 to -58.14], Standard Error of Mean 3.21
Statistical Analysis 11: Comparison: R40 PBO Q2W vs R40 EvoMab Q2W; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -68.31, 95% CI 2-sided [-77.04 to -59.57], Standard Error of Mean 4.42
Statistical Analysis 12: Comparison: R40 PBO QM vs R40 EvoMab QM; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -54.98, 95% CI 2-sided [-65.31 to -44.65], Standard Error of Mean 5.23
Statistical Analysis 13: Comparison: S40 PBO Q2W vs S40 EvoMab Q2W; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -70.56, 95% CI 2-sided [-76.72 to -64.41], Standard Error of Mean 3.12
Statistical Analysis 14: Comparison: S40 PBO QM vs S40 EvoMab QM; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -60.41, 95% CI 2-sided [-69.11 to -51.72], Standard Error of Mean 4.41

2. Primary Outcome: Percent Change From Baseline in LDL-C at the Mean of Weeks 10 and 12
Time Frame: Baseline and Weeks 10 and 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | A10 PBO Q2W | A10 PBO QM | A10 EZE (Q2W) | A10 EZE (QM) | A10 EvoMab Q2W | A10 EvoMab QM | A80 PBO Q2W | A80 PBO QM | A80 EZE (Q2W) | A80 EZE (QM) | A80 EvoMab Q2W | A80 EvoMab QM | R5 PBO Q2W | R5 PBO QM | R5 EvoMab Q2W | R5 EvoMab QM | R40 PBO Q2W | R40 PBO QM | R40 EvoMab Q2W | R40 EvoMab QM | S40 PBO Q2W | S40 PBO QM | S40 EvoMab Q2W | S40 EvoMab QM
Number analyzed (Participants) | 56 | 55 | 56 | 55 | 110 | 110 | 55 | 55 | 56 | 54 | 109 | 110 | 58 | 57 | 113 | 115 | 56 | 55 | 111 | 112 | 56 | 55 | 112 | 115
percent change | 8.54 (2.24) | 0.35 (2.60) | -23.88 (2.34) | -18.98 (2.57) | -61.41 (1.61) | -62.47 (1.83) | 13.12 (3.99) | 9.76 (3.39) | -16.85 (3.88) | -21.25 (3.42) | -61.80 (2.77) | -65.05 (2.42) | 7.55 (2.39) | 2.79 (2.50) | -59.33 (1.74) | -63.79 (1.76) | 6.57 (3.11) | -0.02 (3.51) | -59.08 (2.23) | -62.94 (2.44) | 3.26 (3.40) | 6.00 (4.80) | -66.17 (2.93) | -62.45 (3.85)
Statistical Analysis 1: Comparison: A10 PBO Q2W vs A10 EvoMab Q2W; The null hypothesis was that there was no difference in the percent change from Baseline in the average value of LDL-C at Weeks 10 and 12 between evolocumab and placebo, and the alternative hypothesis was that a mean difference did exist; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -69.95, 95% CI 2-sided [-75.38 to -64.51], Standard Error of Mean 2.76
Statistical Analysis 2: Comparison: A10 PBO QM vs A10 EvoMab QM; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -62.82, 95% CI 2-sided [-69.06 to -56.57], Standard Error of Mean 3.17
Statistical Analysis 3: Comparison: A10 EZE (Q2W) vs A10 EvoMab Q2W; The null hypothesis was that there was no difference in the percent change from Baseline in the average value of LDL-C at Weeks 10 and 12 between evolocumab and ezetimibe, and the alternative hypothesis was that a mean difference did exist; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -37.53, 95% CI 2-sided [-43.03 to -32.03], Standard Error of Mean 2.79
Statistical Analysis 4: Comparison: A10 EZE (QM) vs A10 EvoMab QM; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -43.49, 95% CI 2-sided [-49.70 to -37.28], Standard Error of Mean 3.15
Statistical Analysis 5: Comparison: A80 PBO Q2W vs A80 EvoMab Q2W; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -74.92, 95% CI 2-sided [-84.49 to -65.35], Standard Error of Mean 4.85
Statistical Analysis 6: Comparison: A80 PBO QM vs A80 EvoMab QM; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -74.81, 95% CI 2-sided [-83.00 to -66.62], Standard Error of Mean 4.15
Statistical Analysis 7: Comparison: A80 EZE (Q2W) vs A80 EvoMab Q2W; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -44.95, 95% CI 2-sided [-54.32 to -35.57], Standard Error of Mean 4.75
Statistical Analysis 8: Comparison: A80 EZE (QM) vs A80 EvoMab QM; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -43.81, 95% CI 2-sided [-52.06 to -35.55], Standard Error of Mean 4.19
Statistical Analysis 9: Comparison: R5 PBO Q2W vs R5 EvoMab Q2W; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -66.88, 95% CI 2-sided [-72.67 to -61.08], Standard Error of Mean 2.93
Statistical Analysis 10: Comparison: R5 PBO QM vs R5 EvoMab QM; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -66.58, 95% CI 2-sided [-72.60 to -60.56], Standard Error of Mean 3.05
Statistical Analysis 11: Comparison: R40 PBO Q2W vs R40 EvoMab Q2W; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -65.66, 95% CI 2-sided [-73.19 to -58.12], Standard Error of Mean 3.81
Statistical Analysis 12: Comparison: R40 PBO QM vs R40 EvoMab QM; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -62.91, 95% CI 2-sided [-71.37 to -54.46], Standard Error of Mean 4.27
Statistical Analysis 13: Comparison: S40 PBO Q2W vs S40 EvoMab Q2W; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -69.43, 95% CI 2-sided [-74.86 to -64.01], Standard Error of Mean 2.74
Statistical Analysis 14: Comparison: S40 PBO QM vs S40 EvoMab QM; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -68.45, 95% CI 2-sided [-76.68 to -60.22], Standard Error of Mean 4.17

3. Secondary Outcome: Change From Baseline in LDL-C at at the Mean of Weeks 10 and 12
Time Frame: Baseline and Weeks 10 and 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | A10 PBO Q2W | A10 PBO QM | A10 EZE (Q2W) | A10 EZE (QM) | A10 EvoMab Q2W | A10 EvoMab QM | A80 PBO Q2W | A80 PBO QM | A80 EZE (Q2W) | A80 EZE (QM) | A80 EvoMab Q2W | A80 EvoMab QM | R5 PBO Q2W | R5 PBO QM | R5 EvoMab Q2W | R5 EvoMab QM | R40 PBO Q2W | R40 PBO QM | R40 EvoMab Q2W | R40 EvoMab QM | S40 PBO Q2W | S40 PBO QM | S40 EvoMab Q2W | S40 EvoMab QM
Number analyzed (Participants) | 56 | 55 | 56 | 55 | 110 | 110 | 55 | 55 | 56 | 54 | 109 | 110 | 58 | 57 | 113 | 115 | 56 | 55 | 111 | 112 | 56 | 55 | 112 | 115
mg/dL | 6.8 (3.7) | -0.4 (4.4) | -32.4 (3.8) | -25.1 (4.3) | -76.8 (2.7) | -80.1 (3.1) | 11.0 (5.0) | 5.5 (3.7) | -13.0 (4.9) | -21.3 (3.7) | -58.8 (3.5) | -60.1 (2.6) | 6.5 (3.5) | 0.1 (4.2) | -68.9 (2.5) | -77.8 (3.0) | 3.4 (3.0) | -4.8 (4.2) | -52.3 (2.2) | -55.3 (2.9) | -5.7 (5.2) | 1.7 (6.5) | -83.8 (4.5) | -78.4 (5.1)
Statistical Analysis 1: Comparison: A10 PBO Q2W vs A10 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -83.6, 95% CI 2-sided [-92.6 to -74.6], Standard Error of Mean 4.5
Statistical Analysis 2: Comparison: A10 PBO QM vs A10 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -79.7, 95% CI 2-sided [-90.2 to -69.2], Standard Error of Mean 5.3
Statistical Analysis 3: Comparison: A10 EZE (Q2W) vs A10 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -44.4, 95% CI 2-sided [-53.4 to -35.3], Standard Error of Mean 4.4
Statistical Analysis 4: Comparison: A10 EZE (QM) vs A10 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -55.0, 95% CI 2-sided [-65.4 to -44.6], Standard Error of Mean 5.3
Statistical Analysis 5: Comparison: A80 PBO Q2W vs A80 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -69.9, 95% CI 2-sided [-81.9 to -57.8], Standard Error of Mean 6.1
Statistical Analysis 6: Comparison: A80 PBO QM vs A80 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -65.6, 95% CI 2-sided [-74.5 to -56.7], Standard Error of Mean 4.5
Statistical Analysis 7: Comparison: A80 EZE (Q2W) vs A80 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -45.8, 95% CI 2-sided [-57.7 to -33.9], Standard Error of Mean 6.0
Statistical Analysis 8: Comparison: A80 EZE (QM) vs A80 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -38.8, 95% CI 2-sided [-47.8 to -29.9], Standard Error of Mean 4.5
Statistical Analysis 9: Comparison: R5 PBO Q2W vs R5 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -75.4, 95% CI 2-sided [-83.9 to -67.0], Standard Error of Mean 4.3
Statistical Analysis 10: Comparison: R5 PBO QM vs R5 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -77.9, 95% CI 2-sided [-88.0 to -67.8], Standard Error of Mean 5.1
Statistical Analysis 11: Comparison: R40 PBO Q2W vs R40 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -55.8, 95% CI 2-sided [-63.1 to -48.4], Standard Error of Mean 3.7
Statistical Analysis 12: Comparison: R40 PBO QM vs R40 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -50.6, 95% CI 2-sided [-60.6 to -40.6], Standard Error of Mean 5.1
Statistical Analysis 13: Comparison: S40 PBO Q2W vs S40 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -78.1, 95% CI 2-sided [-86.2 to -70.0], Standard Error of Mean 4.1
Statistical Analysis 14: Comparison: S40 PBO QM vs S40 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -80.1, 95% CI 2-sided [-91.7 to -68.6], Standard Error of Mean 5.8

4. Secondary Outcome: Change From Baseline in LDL-C at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | A10 PBO Q2W | A10 PBO QM | A10 EZE (Q2W) | A10 EZE (QM) | A10 EvoMab Q2W | A10 EvoMab QM | A80 PBO Q2W | A80 PBO QM | A80 EZE (Q2W) | A80 EZE (QM) | A80 EvoMab Q2W | A80 EvoMab QM | R5 PBO Q2W | R5 PBO QM | R5 EvoMab Q2W | R5 EvoMab QM | R40 PBO Q2W | R40 PBO QM | R40 EvoMab Q2W | R40 EvoMab QM | S40 PBO Q2W | S40 PBO QM | S40 EvoMab Q2W | S40 EvoMab QM
Number analyzed (Participants) | 56 | 55 | 56 | 55 | 110 | 110 | 55 | 55 | 56 | 54 | 109 | 110 | 58 | 57 | 113 | 115 | 56 | 55 | 111 | 112 | 56 | 55 | 112 | 115
mg/dL | 8.6 (4.0) | 0.8 (4.5) | -30.1 (4.1) | -23.3 (4.5) | -77.0 (2.9) | -75.1 (3.2) | 12.7 (5.3) | 7.0 (4.1) | -9.9 (5.2) | -19.5 (4.1) | -59.0 (3.7) | -54.8 (2.9) | 7.8 (3.8) | 2.4 (4.4) | -69.2 (2.7) | -73.3 (3.1) | 5.1 (3.2) | -2.0 (4.7) | -52.1 (2.3) | -46.7 (3.3) | -4.5 (5.3) | -0.6 (6.6) | -83.5 (4.6) | -72.5 (5.2)
Statistical Analysis 1: Comparison: A10 PBO Q2W vs A10 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -85.5, 95% CI 2-sided [-95.2 to -75.9], Standard Error of Mean 4.9
Statistical Analysis 2: Comparison: A10 PBO QM vs A10 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -75.8, 95% CI 2-sided [-86.8 to -64.9], Standard Error of Mean 5.5
Statistical Analysis 3: Comparison: A10 EZE (Q2W) vs A10 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -46.8, 95% CI 2-sided [-56.6 to -37.1], Standard Error of Mean 4.9
Statistical Analysis 4: Comparison: A10 EZE (QM) vs A10 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -51.7, 95% CI 2-sided [-62.6 to -40.9], Standard Error of Mean 5.5
Statistical Analysis 5: Comparison: A80 PBO Q2W vs A80 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -71.7, 95% CI 2-sided [-84.4 to -59.0], Standard Error of Mean 6.4
Statistical Analysis 6: Comparison: A80 PBO QM vs A80 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -61.8, 95% CI 2-sided [-71.6 to -52.0], Standard Error of Mean 5.0
Statistical Analysis 7: Comparison: A80 EZE (Q2W) vs A80 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -49.0, 95% CI 2-sided [-61.5 to -36.6], Standard Error of Mean 6.3
Statistical Analysis 8: Comparison: A80 EZE (QM) vs A80 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -35.3, 95% CI 2-sided [-45.2 to -25.5], Standard Error of Mean 5.0
Statistical Analysis 9: Comparison: R5 PBO Q2W vs R5 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -77.1, 95% CI 2-sided [-86.2 to -67.9], Standard Error of Mean 4.6
Statistical Analysis 10: Comparison: R5 PBO QM vs R5 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -75.8, 95% CI 2-sided [-86.3 to -65.3], Standard Error of Mean 5.3
Statistical Analysis 11: Comparison: R40 PBO Q2W vs R40 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -57.2, 95% CI 2-sided [-65.1 to -49.4], Standard Error of Mean 4.0
Statistical Analysis 12: Comparison: R40 PBO QM vs R40 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -44.6, 95% CI 2-sided [-55.9 to -33.4], Standard Error of Mean 5.7
Statistical Analysis 13: Comparison: S40 PBO Q2W vs S40 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -79.0, 95% CI 2-sided [-87.5 to -70.4], Standard Error of Mean 4.3
Statistical Analysis 14: Comparison: S40 PBO QM vs S40 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -71.9, 95% CI 2-sided [-83.8 to -60.0], Standard Error of Mean 6.0

5. Secondary Outcome: Percent Change From Baseline in Non-High-Density Lipoprotein Cholesterol (Non-HDL-C) at the Mean of Weeks 10 and 12
Time Frame: Baseline and Weeks 10 and 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | A10 PBO Q2W | A10 PBO QM | A10 EZE (Q2W) | A10 EZE (QM) | A10 EvoMab Q2W | A10 EvoMab QM | A80 PBO Q2W | A80 PBO QM | A80 EZE (Q2W) | A80 EZE (QM) | A80 EvoMab Q2W | A80 EvoMab QM | R5 PBO Q2W | R5 PBO QM | R5 EvoMab Q2W | R5 EvoMab QM | R40 PBO Q2W | R40 PBO QM | R40 EvoMab Q2W | R40 EvoMab QM | S40 PBO Q2W | S40 PBO QM | S40 EvoMab Q2W | S40 EvoMab QM
Number analyzed (Participants) | 56 | 55 | 56 | 55 | 110 | 110 | 55 | 55 | 56 | 54 | 109 | 110 | 58 | 57 | 113 | 115 | 56 | 55 | 111 | 112 | 56 | 55 | 112 | 115
percent change | 6.80 (2.07) | 1.28 (2.44) | -20.71 (2.15) | -16.56 (2.41) | -53.48 (1.48) | -56.09 (1.71) | 10.74 (3.59) | 8.45 (3.13) | -16.19 (3.49) | -18.79 (3.16) | -54.44 (2.49) | -56.31 (2.23) | 7.02 (2.11) | 3.73 (2.32) | -52.59 (1.54) | -55.47 (1.64) | 6.19 (2.61) | 1.58 (2.90) | -52.08 (1.88) | -55.72 (2.01) | 0.74 (3.23) | 6.81 (4.35) | -59.33 (2.79) | -56.01 (3.49)
Statistical Analysis 1: Comparison: A10 PBO Q2W vs A10 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -60.28, 95% CI 2-sided [-65.29 to -55.27], Standard Error of Mean 2.54
Statistical Analysis 2: Comparison: A10 PBO QM vs A10 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -57.37, 95% CI 2-sided [-63.23 to -51.51], Standard Error of Mean 2.97
Statistical Analysis 3: Comparison: A10 EZE (Q2W) vs A10 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -32.77, 95% CI 2-sided [-37.84 to -27.70], Standard Error of Mean 2.57
Statistical Analysis 4: Comparison: A10 EZE (QM) vs A10 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -39.53, 95% CI 2-sided [-45.34 to -33.71], Standard Error of Mean 2.95
Statistical Analysis 5: Comparison: A80 PBO Q2W vs A80 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -65.17, 95% CI 2-sided [-73.78 to -56.56], Standard Error of Mean 4.37
Statistical Analysis 6: Comparison: A80 PBO QM vs A80 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -64.76, 95% CI 2-sided [-72.32 to -57.19], Standard Error of Mean 3.84
Statistical Analysis 7: Comparison: A80 EZE (Q2W) vs A80 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -38.25, 95% CI 2-sided [-46.68 to -29.81], Standard Error of Mean 4.28
Statistical Analysis 8: Comparison: A80 EZE (QM) vs A80 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -37.52, 95% CI 2-sided [-45.15 to -29.90], Standard Error of Mean 3.87
Statistical Analysis 9: Comparison: R5 PBO Q2W vs R5 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -59.61, 95% CI 2-sided [-64.73 to -54.48], Standard Error of Mean 2.60
Statistical Analysis 10: Comparison: R5 PBO QM vs R5 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -59.20, 95% CI 2-sided [-64.80 to -53.60], Standard Error of Mean 2.83
Statistical Analysis 11: Comparison: R40 PBO Q2W vs R40 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -58.27, 95% CI 2-sided [-64.60 to -51.94], Standard Error of Mean 3.20
Statistical Analysis 12: Comparison: R40 PBO QM vs R40 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -57.31, 95% CI 2-sided [-64.29 to -50.32], Standard Error of Mean 3.53
Statistical Analysis 13: Comparison: S40 PBO Q2W vs S40 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -60.06, 95% CI 2-sided [-65.18 to -54.94], Standard Error of Mean 2.59
Statistical Analysis 14: Comparison: S40 PBO QM vs S40 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -62.82, 95% CI 2-sided [-70.22 to -55.42], Standard Error of Mean 3.75

6. Secondary Outcome: Percent Change From Baseline in Non-HDL-C at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | A10 PBO Q2W | A10 PBO QM | A10 EZE (Q2W) | A10 EZE (QM) | A10 EvoMab Q2W | A10 EvoMab QM | A80 PBO Q2W | A80 PBO QM | A80 EZE (Q2W) | A80 EZE (QM) | A80 EvoMab Q2W | A80 EvoMab QM | R5 PBO Q2W | R5 PBO QM | R5 EvoMab Q2W | R5 EvoMab QM | R40 PBO Q2W | R40 PBO QM | R40 EvoMab Q2W | R40 EvoMab QM | S40 PBO Q2W | S40 PBO QM | S40 EvoMab Q2W | S40 EvoMab QM
Number analyzed (Participants) | 56 | 55 | 56 | 55 | 110 | 110 | 55 | 55 | 56 | 54 | 109 | 110 | 58 | 57 | 113 | 115 | 56 | 55 | 111 | 112 | 56 | 55 | 112 | 115
percent change | 8.25 (2.32) | 2.43 (2.69) | -18.27 (2.40) | -14.78 (2.65) | -53.39 (1.66) | -52.20 (1.90) | 11.79 (3.87) | 9.95 (3.51) | -14.34 (3.75) | -17.26 (3.52) | -54.84 (2.66) | -50.05 (2.50) | 7.92 (2.40) | 5.85 (2.42) | -52.04 (1.74) | -51.57 (1.72) | 8.61 (3.04) | 3.35 (3.53) | -50.97 (2.18) | -46.42 (2.45) | 1.89 (3.38) | 5.66 (4.53) | -59.02 (2.87) | -50.96 (3.60)
Statistical Analysis 1: Comparison: A10 PBO Q2W vs A10 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -61.64, 95% CI 2-sided [-67.25 to -56.03], Standard Error of Mean 2.84
Statistical Analysis 2: Comparison: A10 PBO QM vs A10 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -54.93, 95% CI 2-sided [-61.40 to -48.46], Standard Error of Mean 3.28
Statistical Analysis 3: Comparison: A10 EZE (Q2W) vs A10 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -35.11, 95% CI 2-sided [-40.79 to -29.44], Standard Error of Mean 2.88
Statistical Analysis 4: Comparison: A10 EZE (QM) vs A10 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -37.72, 95% CI 2-sided [-44.15 to -31.30], Standard Error of Mean 3.26
Statistical Analysis 5: Comparison: A80 PBO Q2W vs A80 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -66.64, 95% CI 2-sided [-75.88 to -57.39], Standard Error of Mean 4.69
Statistical Analysis 6: Comparison: A80 PBO QM vs A80 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -60.01, 95% CI 2-sided [-68.49 to -51.52], Standard Error of Mean 4.30
Statistical Analysis 7: Comparison: A80 EZE (Q2W) vs A80 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -40.51, 95% CI 2-sided [-49.55 to -31.47], Standard Error of Mean 4.59
Statistical Analysis 8: Comparison: A80 EZE (QM) vs A80 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -32.79, 95% CI 2-sided [-41.30 to -24.28], Standard Error of Mean 4.32
Statistical Analysis 9: Comparison: R5 PBO Q2W vs R5 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -59.96, 95% CI 2-sided [-65.78 to -54.13], Standard Error of Mean 2.95
Statistical Analysis 10: Comparison: R5 PBO QM vs R5 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -57.42, 95% CI 2-sided [-63.27 to -51.57], Standard Error of Mean 2.96
Statistical Analysis 11: Comparison: R40 PBO Q2W vs R40 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -59.58, 95% CI 2-sided [-66.95 to -52.21], Standard Error of Mean 3.73
Statistical Analysis 12: Comparison: R40 PBO QM vs R40 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -49.76, 95% CI 2-sided [-58.26 to -41.27], Standard Error of Mean 4.30
Statistical Analysis 13: Comparison: S40 PBO Q2W vs S40 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -60.91, 95% CI 2-sided [-66.57 to -55.24], Standard Error of Mean 2.87
Statistical Analysis 14: Comparison: S40 PBO QM vs S40 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -56.63, 95% CI 2-sided [-64.63 to -48.62], Standard Error of Mean 4.06

7. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B at the Mean of Weeks 10 and 12
Time Frame: Baseline and Weeks 10 and 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | A10 PBO Q2W | A10 PBO QM | A10 EZE (Q2W) | A10 EZE (QM) | A10 EvoMab Q2W | A10 EvoMab QM | A80 PBO Q2W | A80 PBO QM | A80 EZE (Q2W) | A80 EZE (QM) | A80 EvoMab Q2W | A80 EvoMab QM | R5 PBO Q2W | R5 PBO QM | R5 EvoMab Q2W | R5 EvoMab QM | R40 PBO Q2W | R40 PBO QM | R40 EvoMab Q2W | R40 EvoMab QM | S40 PBO Q2W | S40 PBO QM | S40 EvoMab Q2W | S40 EvoMab QM
Number analyzed (Participants) | 56 | 55 | 56 | 55 | 110 | 110 | 55 | 55 | 56 | 54 | 109 | 110 | 58 | 57 | 113 | 115 | 56 | 55 | 111 | 112 | 56 | 55 | 112 | 115
percent change | 7.55 (1.89) | 0.81 (2.19) | -17.29 (2.00) | -11.43 (2.20) | -50.95 (1.38) | -51.44 (1.52) | 10.20 (3.02) | 5.48 (2.83) | -14.22 (2.98) | -13.62 (2.87) | -49.14 (2.13) | -53.26 (2.02) | 5.07 (1.97) | 2.54 (1.89) | -49.79 (1.46) | -53.59 (1.32) | 3.71 (2.46) | 1.98 (2.57) | -47.07 (1.76) | -52.95 (1.76) | -0.31 (3.02) | 2.49 (4.67) | -55.65 (2.63) | -54.37 (3.93)
Statistical Analysis 1: Comparison: A10 PBO Q2W vs A10 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -58.49, 95% CI 2-sided [-63.10 to -53.89], Standard Error of Mean 2.34
Statistical Analysis 2: Comparison: A10 PBO QM vs A10 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -52.25, 95% CI 2-sided [-57.49 to -47.01], Standard Error of Mean 2.66
Statistical Analysis 3: Comparison: A10 EZE (Q2W) vs A10 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -33.66, 95% CI 2-sided [-38.33 to -28.98], Standard Error of Mean 2.37
Statistical Analysis 4: Comparison: A10 EZE (QM) vs A10 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -40.01, 95% CI 2-sided [-45.27 to -34.74], Standard Error of Mean 2.67
Statistical Analysis 5: Comparison: A80 PBO Q2W vs A80 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -59.34, 95% CI 2-sided [-66.61 to -52.07], Standard Error of Mean 3.69
Statistical Analysis 6: Comparison: A80 PBO QM vs A80 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -58.74, 95% CI 2-sided [-65.56 to -51.93], Standard Error of Mean 3.46
Statistical Analysis 7: Comparison: A80 EZE (Q2W) vs A80 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -34.92, 95% CI 2-sided [-42.09 to -27.75], Standard Error of Mean 3.64
Statistical Analysis 8: Comparison: A80 EZE (QM) vs A80 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -39.64, 95% CI 2-sided [-46.57 to -32.71], Standard Error of Mean 3.52
Statistical Analysis 9: Comparison: R5 PBO Q2W vs R5 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -54.86, 95% CI 2-sided [-59.66 to -50.05], Standard Error of Mean 2.43
Statistical Analysis 10: Comparison: R5 PBO QM vs R5 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -56.14, 95% CI 2-sided [-60.66 to -51.61], Standard Error of Mean 2.29
Statistical Analysis 11: Comparison: R40 PBO Q2W vs R40 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -50.78, 95% CI 2-sided [-56.72 to -44.83], Standard Error of Mean 3.01
Statistical Analysis 12: Comparison: R40 PBO QM vs R40 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -54.94, 95% CI 2-sided [-61.11 to -48.76], Standard Error of Mean 3.12
Statistical Analysis 13: Comparison: S40 PBO Q2W vs S40 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -55.34, 95% CI 2-sided [-59.94 to -50.74], Standard Error of Mean 2.33
Statistical Analysis 14: Comparison: S40 PBO QM vs S40 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -56.87, 95% CI 2-sided [-63.27 to -50.46], Standard Error of Mean 3.24

8. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | A10 PBO Q2W | A10 PBO QM | A10 EZE (Q2W) | A10 EZE (QM) | A10 EvoMab Q2W | A10 EvoMab QM | A80 PBO Q2W | A80 PBO QM | A80 EZE (Q2W) | A80 EZE (QM) | A80 EvoMab Q2W | A80 EvoMab QM | R5 PBO Q2W | R5 PBO QM | R5 EvoMab Q2W | R5 EvoMab QM | R40 PBO Q2W | R40 PBO QM | R40 EvoMab Q2W | R40 EvoMab QM | S40 PBO Q2W | S40 PBO QM | S40 EvoMab Q2W | S40 EvoMab QM
Number analyzed (Participants) | 56 | 55 | 56 | 55 | 110 | 110 | 55 | 55 | 56 | 54 | 109 | 110 | 58 | 57 | 113 | 115 | 56 | 55 | 111 | 112 | 56 | 55 | 112 | 115
percent change | 7.89 (2.16) | 0.21 (2.43) | -15.98 (2.26) | -10.95 (2.44) | -50.90 (1.56) | -47.15 (1.70) | 11.64 (3.28) | 6.54 (3.22) | -12.31 (3.20) | -12.16 (3.24) | -49.77 (2.28) | -46.47 (2.31) | 6.35 (2.10) | 4.63 (2.11) | -50.15 (1.54) | -48.58 (1.49) | 4.91 (2.71) | 3.24 (3.13) | -45.61 (1.93) | -43.71 (2.13) | 0.35 (3.17) | 3.57 (4.74) | -55.95 (2.72) | -49.16 (3.97)
Statistical Analysis 1: Comparison: A10 PBO Q2W vs A10 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -58.79, 95% CI 2-sided [-64.03 to -53.55], Standard Error of Mean 2.66
Statistical Analysis 2: Comparison: A10 PBO QM vs A10 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -47.36, 95% CI 2-sided [-53.20 to -41.52], Standard Error of Mean 2.96
Statistical Analysis 3: Comparison: A10 EZE (Q2W) vs A10 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -34.92, 95% CI 2-sided [-40.23 to -29.60], Standard Error of Mean 2.69
Statistical Analysis 4: Comparison: A10 EZE (QM) vs A10 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -36.21, 95% CI 2-sided [-42.06 to -30.35], Standard Error of Mean 2.97
Statistical Analysis 5: Comparison: A80 PBO Q2W vs A80 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -61.40, 95% CI 2-sided [-69.27 to -53.54], Standard Error of Mean 3.99
Statistical Analysis 6: Comparison: A80 PBO QM vs A80 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -53.01, 95% CI 2-sided [-60.77 to -45.25], Standard Error of Mean 3.93
Statistical Analysis 7: Comparison: A80 EZE (Q2W) vs A80 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -37.45, 95% CI 2-sided [-45.17 to -29.74], Standard Error of Mean 3.91
Statistical Analysis 8: Comparison: A80 EZE (QM) vs A80 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -34.31, 95% CI 2-sided [-42.15 to -26.47], Standard Error of Mean 3.98
Statistical Analysis 9: Comparison: R5 PBO Q2W vs R5 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -56.50, 95% CI 2-sided [-61.60 to -51.40], Standard Error of Mean 2.58
Statistical Analysis 10: Comparison: R5 PBO QM vs R5 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -53.21, 95% CI 2-sided [-58.29 to -48.13], Standard Error of Mean 2.57
Statistical Analysis 11: Comparison: R40 PBO Q2W vs R40 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -50.52, 95% CI 2-sided [-57.06 to -43.99], Standard Error of Mean 3.31
Statistical Analysis 12: Comparison: R40 PBO QM vs R40 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -46.95, 95% CI 2-sided [-54.43 to -39.47], Standard Error of Mean 3.78
Statistical Analysis 13: Comparison: S40 PBO Q2W vs S40 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -56.30, 95% CI 2-sided [-61.47 to -51.14], Standard Error of Mean 2.61
Statistical Analysis 14: Comparison: S40 PBO QM vs S40 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -52.73, 95% CI 2-sided [-59.40 to -46.06], Standard Error of Mean 3.38

9. Secondary Outcome: Percent Change From Baseline in the Total Cholesterol/HDL-C Ratio at the Mean of Weeks 10 and 12
Time Frame: Baseline and Weeks 10 and 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | A10 PBO Q2W | A10 PBO QM | A10 EZE (Q2W) | A10 EZE (QM) | A10 EvoMab Q2W | A10 EvoMab QM | A80 PBO Q2W | A80 PBO QM | A80 EZE (Q2W) | A80 EZE (QM) | A80 EvoMab Q2W | A80 EvoMab QM | R5 PBO Q2W | R5 PBO QM | R5 EvoMab Q2W | R5 EvoMab QM | R40 PBO Q2W | R40 PBO QM | R40 EvoMab Q2W | R40 EvoMab QM | S40 PBO Q2W | S40 PBO QM | S40 EvoMab Q2W | S40 EvoMab QM
Number analyzed (Participants) | 56 | 55 | 56 | 55 | 110 | 110 | 55 | 55 | 56 | 54 | 109 | 110 | 58 | 57 | 113 | 115 | 56 | 55 | 111 | 112 | 56 | 55 | 112 | 115
percent change | 5.96 (1.76) | 2.24 (2.11) | -14.39 (1.83) | -10.86 (2.08) | -40.44 (1.26) | -42.45 (1.48) | 4.26 (2.59) | 6.42 (2.34) | -11.92 (2.52) | -12.25 (2.35) | -40.22 (1.80) | -40.43 (1.66) | 5.41 (1.96) | 5.02 (2.25) | -39.33 (1.43) | -42.00 (1.59) | 4.55 (1.98) | 1.71 (2.36) | -36.04 (1.42) | -38.62 (1.64) | -0.14 (2.79) | 5.45 (3.50) | -47.20 (2.37) | -43.17 (2.85)
Statistical Analysis 1: Comparison: A10 PBO Q2W vs A10 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -46.41, 95% CI 2-sided [-50.66 to -42.15], Standard Error of Mean 2.16
Statistical Analysis 2: Comparison: A10 PBO QM vs A10 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -44.69, 95% CI 2-sided [-49.75 to -39.63], Standard Error of Mean 2.57
Statistical Analysis 3: Comparison: A10 EZE (Q2W) vs A10 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -26.06, 95% CI 2-sided [-30.36 to -21.75], Standard Error of Mean 2.19
Statistical Analysis 4: Comparison: A10 EZE (QM) vs A10 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -31.59, 95% CI 2-sided [-36.61 to -26.57], Standard Error of Mean 2.55
Statistical Analysis 5: Comparison: A80 PBO Q2W vs A80 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -44.48, 95% CI 2-sided [-50.69 to -38.27], Standard Error of Mean 3.15
Statistical Analysis 6: Comparison: A80 PBO QM vs A80 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -46.85, 95% CI 2-sided [-52.48 to -41.21], Standard Error of Mean 2.86
Statistical Analysis 7: Comparison: A80 EZE (Q2W) vs A80 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -28.30, 95% CI 2-sided [-34.39 to -22.21], Standard Error of Mean 3.09
Statistical Analysis 8: Comparison: A80 EZE (QM) vs A80 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -28.18, 95% CI 2-sided [-33.86 to -22.50], Standard Error of Mean 2.88
Statistical Analysis 9: Comparison: R5 PBO Q2W vs R5 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -44.73, 95% CI 2-sided [-49.50 to -39.97], Standard Error of Mean 2.41
Statistical Analysis 10: Comparison: R5 PBO QM vs R5 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -47.01, 95% CI 2-sided [-52.46 to -41.57], Standard Error of Mean 2.75
Statistical Analysis 11: Comparison: R40 PBO Q2W vs R40 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -40.59, 95% CI 2-sided [-45.38 to -35.79], Standard Error of Mean 2.43
Statistical Analysis 12: Comparison: R40 PBO QM vs R40 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -40.33, 95% CI 2-sided [-46.00 to -34.66], Standard Error of Mean 2.87
Statistical Analysis 13: Comparison: S40 PBO Q2W vs S40 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -47.05, 95% CI 2-sided [-51.76 to -42.35], Standard Error of Mean 2.38
Statistical Analysis 14: Comparison: S40 PBO QM vs S40 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -48.62, 95% CI 2-sided [-54.27 to -42.98], Standard Error of Mean 2.86

10. Secondary Outcome: Percent Change From Baseline in the Total Cholesterol/HDL-C Ratio at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | A10 PBO Q2W | A10 PBO QM | A10 EZE (Q2W) | A10 EZE (QM) | A10 EvoMab Q2W | A10 EvoMab QM | A80 PBO Q2W | A80 PBO QM | A80 EZE (Q2W) | A80 EZE (QM) | A80 EvoMab Q2W | A80 EvoMab QM | R5 PBO Q2W | R5 PBO QM | R5 EvoMab Q2W | R5 EvoMab QM | R40 PBO Q2W | R40 PBO QM | R40 EvoMab Q2W | R40 EvoMab QM | S40 PBO Q2W | S40 PBO QM | S40 EvoMab Q2W | S40 EvoMab QM
Number analyzed (Participants) | 56 | 55 | 56 | 55 | 110 | 110 | 55 | 55 | 56 | 54 | 109 | 110 | 58 | 57 | 113 | 115 | 56 | 55 | 111 | 112 | 56 | 55 | 112 | 115
percent change | 6.09 (2.02) | 2.80 (2.31) | -12.14 (2.10) | -9.85 (2.28) | -40.74 (1.45) | -40.07 (1.63) | 4.31 (2.75) | 6.18 (2.73) | -10.53 (2.66) | -11.06 (2.73) | -40.79 (1.89) | -36.25 (1.94) | 4.68 (2.28) | 6.07 (2.36) | -38.57 (1.64) | -39.26 (1.68) | 5.96 (2.28) | 2.69 (2.80) | -35.17 (1.63) | -32.30 (1.94) | -0.20 (2.81) | 5.13 (3.62) | -47.24 (2.38) | -39.47 (2.92)
Statistical Analysis 1: Comparison: A10 PBO Q2W vs A10 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -46.83, 95% CI 2-sided [-51.73 to -41.94], Standard Error of Mean 2.48
Statistical Analysis 2: Comparison: A10 PBO QM vs A10 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -42.86, 95% CI 2-sided [-48.43 to -37.30], Standard Error of Mean 2.82
Statistical Analysis 3: Comparison: A10 EZE (Q2W) vs A10 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -28.60, 95% CI 2-sided [-33.56 to -23.65], Standard Error of Mean 2.51
Statistical Analysis 4: Comparison: A10 EZE (QM) vs A10 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -30.22, 95% CI 2-sided [-35.74 to -24.70], Standard Error of Mean 2.80
Statistical Analysis 5: Comparison: A80 PBO Q2W vs A80 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -45.10, 95% CI 2-sided [-51.66 to -38.54], Standard Error of Mean 3.33
Statistical Analysis 6: Comparison: A80 PBO QM vs A80 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -42.43, 95% CI 2-sided [-49.01 to -35.85], Standard Error of Mean 3.34
Statistical Analysis 7: Comparison: A80 EZE (Q2W) vs A80 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -30.26, 95% CI 2-sided [-36.68 to -23.84], Standard Error of Mean 3.26
Statistical Analysis 8: Comparison: A80 EZE (QM) vs A80 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -25.19, 95% CI 2-sided [-31.79 to -18.59], Standard Error of Mean 3.35
Statistical Analysis 9: Comparison: R5 PBO Q2W vs R5 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -43.25, 95% CI 2-sided [-48.77 to -37.74], Standard Error of Mean 2.79
Statistical Analysis 10: Comparison: R5 PBO QM vs R5 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -45.33, 95% CI 2-sided [-51.04 to -39.61], Standard Error of Mean 2.89
Statistical Analysis 11: Comparison: R40 PBO Q2W vs R40 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -41.13, 95% CI 2-sided [-46.65 to -35.61], Standard Error of Mean 2.79
Statistical Analysis 12: Comparison: R40 PBO QM vs R40 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -34.99, 95% CI 2-sided [-41.72 to -28.25], Standard Error of Mean 3.41
Statistical Analysis 13: Comparison: S40 PBO Q2W vs S40 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -47.04, 95% CI 2-sided [-51.83 to -42.25], Standard Error of Mean 2.43
Statistical Analysis 14: Comparison: S40 PBO QM vs S40 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -44.60, 95% CI 2-sided [-50.67 to -38.54], Standard Error of Mean 3.07

11. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B/Apolipoprotein A1 Ratio at the Mean of Weeks 10 and 12
Time Frame: Baseline and Weeks 10 and 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | A10 PBO Q2W | A10 PBO QM | A10 EZE (Q2W) | A10 EZE (QM) | A10 EvoMab Q2W | A10 EvoMab QM | A80 PBO Q2W | A80 PBO QM | A80 EZE (Q2W) | A80 EZE (QM) | A80 EvoMab Q2W | A80 EvoMab QM | R5 PBO Q2W | R5 PBO QM | R5 EvoMab Q2W | R5 EvoMab QM | R40 PBO Q2W | R40 PBO QM | R40 EvoMab Q2W | R40 EvoMab QM | S40 PBO Q2W | S40 PBO QM | S40 EvoMab Q2W | S40 EvoMab QM
Number analyzed (Participants) | 56 | 55 | 56 | 55 | 110 | 110 | 55 | 55 | 56 | 54 | 109 | 110 | 58 | 57 | 113 | 115 | 56 | 55 | 111 | 112 | 56 | 55 | 112 | 115
percent change | 6.41 (2.03) | 0.78 (2.29) | -15.77 (2.14) | -11.47 (2.29) | -53.56 (1.48) | -53.33 (1.58) | 4.48 (3.04) | 5.79 (2.79) | -15.17 (2.99) | -12.91 (2.80) | -52.43 (2.14) | -56.20 (1.98) | 2.82 (2.26) | 2.58 (2.05) | -52.46 (1.67) | -56.66 (1.43) | 2.17 (2.56) | 2.60 (2.97) | -48.47 (1.83) | -54.17 (2.04) | -1.00 (3.12) | -1.42 (4.22) | -58.76 (2.73) | -57.47 (3.55)
Statistical Analysis 1: Comparison: A10 PBO Q2W vs A10 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -59.97, 95% CI 2-sided [-64.91 to -55.03], Standard Error of Mean 2.51
Statistical Analysis 2: Comparison: A10 PBO QM vs A10 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -54.11, 95% CI 2-sided [-59.57 to -48.64], Standard Error of Mean 2.77
Statistical Analysis 3: Comparison: A10 EZE (Q2W) vs A10 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -37.79, 95% CI 2-sided [-42.80 to -32.77], Standard Error of Mean 2.54
Statistical Analysis 4: Comparison: A10 EZE (QM) vs A10 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -41.86, 95% CI 2-sided [-47.34 to -36.67], Standard Error of Mean 2.78
Statistical Analysis 5: Comparison: A80 PBO Q2W vs A80 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -56.90, 95% CI 2-sided [-64.22 to -49.59], Standard Error of Mean 3.71
Statistical Analysis 6: Comparison: A80 PBO QM vs A80 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -61.99, 95% CI 2-sided [-68.68 to -55.29], Standard Error of Mean 3.39
Statistical Analysis 7: Comparison: A80 EZE (Q2W) vs A80 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -37.26, 95% CI 2-sided [-44.48 to -30.04], Standard Error of Mean 3.66
Statistical Analysis 8: Comparison: A80 EZE (QM) vs A80 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -43.29, 95% CI 2-sided [-50.07 to -36.51], Standard Error of Mean 3.44
Statistical Analysis 9: Comparison: R5 PBO Q2W vs R5 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -55.29, 95% CI 2-sided [-60.79 to -49.79], Standard Error of Mean 2.78
Statistical Analysis 10: Comparison: R5 PBO QM vs R5 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -59.24, 95% CI 2-sided [-64.16 to -54.32], Standard Error of Mean 2.49
Statistical Analysis 11: Comparison: R40 PBO Q2W vs R40 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -50.63, 95% CI 2-sided [-56.82 to -44.45], Standard Error of Mean 3.13
Statistical Analysis 12: Comparison: R40 PBO QM vs R40 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -56.78, 95% CI 2-sided [-63.91 to -49.64], Standard Error of Mean 3.61
Statistical Analysis 13: Comparison: S40 PBO Q2W vs S40 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -57.75, 95% CI 2-sided [-62.51 to -52.99], Standard Error of Mean 2.41
Statistical Analysis 14: Comparison: S40 PBO QM vs S40 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -56.06, 95% CI 2-sided [-61.85 to -50.27], Standard Error of Mean 2.93

12. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B/Apolipoprotein A1 Ratio at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | A10 PBO Q2W | A10 PBO QM | A10 EZE (Q2W) | A10 EZE (QM) | A10 EvoMab Q2W | A10 EvoMab QM | A80 PBO Q2W | A80 PBO QM | A80 EZE (Q2W) | A80 EZE (QM) | A80 EvoMab Q2W | A80 EvoMab QM | R5 PBO Q2W | R5 PBO QM | R5 EvoMab Q2W | R5 EvoMab QM | R40 PBO Q2W | R40 PBO QM | R40 EvoMab Q2W | R40 EvoMab QM | S40 PBO Q2W | S40 PBO QM | S40 EvoMab Q2W | S40 EvoMab QM
Number analyzed (Participants) | 56 | 55 | 56 | 55 | 110 | 110 | 55 | 55 | 56 | 54 | 109 | 110 | 58 | 57 | 113 | 115 | 56 | 55 | 111 | 112 | 56 | 55 | 112 | 115
percent change | 6.13 (2.20) | -1.21 (2.41) | -14.51 (2.31) | -12.33 (2.41) | -54.17 (1.59) | -49.65 (1.69) | 4.19 (3.25) | 6.50 (3.18) | -13.69 (3.17) | -12.19 (3.17) | -53.59 (2.26) | -50.76 (2.26) | 1.44 (2.30) | 4.00 (2.27) | -52.97 (1.69) | -52.13 (1.60) | 1.64 (2.75) | 3.16 (3.51) | -47.53 (1.96) | -45.65 (2.39) | -1.80 (3.21) | -0.52 (4.29) | -59.53 (2.77) | -52.56 (3.59)
Statistical Analysis 1: Comparison: A10 PBO Q2W vs A10 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -60.29, 95% CI 2-sided [-65.65 to -54.94], Standard Error of Mean 2.71
Statistical Analysis 2: Comparison: A10 PBO QM vs A10 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -48.44, 95% CI 2-sided [-54.23 to -42.65], Standard Error of Mean 2.94
Statistical Analysis 3: Comparison: A10 EZE (Q2W) vs A10 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -39.66, 95% CI 2-sided [-45.09 to -34.23], Standard Error of Mean 2.75
Statistical Analysis 4: Comparison: A10 EZE (QM) vs A10 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -37.32, 95% CI 2-sided [-43.12 to -31.52], Standard Error of Mean 2.94
Statistical Analysis 5: Comparison: A80 PBO Q2W vs A80 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -57.77, 95% CI 2-sided [-65.55 to -49.99], Standard Error of Mean 3.95
Statistical Analysis 6: Comparison: A80 PBO QM vs A80 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -57.26, 95% CI 2-sided [-64.91 to -49.60], Standard Error of Mean 3.88
Statistical Analysis 7: Comparison: A80 EZE (Q2W) vs A80 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -39.90, 95% CI 2-sided [-47.53 to -32.26], Standard Error of Mean 3.87
Statistical Analysis 8: Comparison: A80 EZE (QM) vs A80 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -38.57, 95% CI 2-sided [-46.26 to -30.88], Standard Error of Mean 3.90
Statistical Analysis 9: Comparison: R5 PBO Q2W vs R5 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -54.41, 95% CI 2-sided [-59.99 to -48.82], Standard Error of Mean 2.83
Statistical Analysis 10: Comparison: R5 PBO QM vs R5 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -56.13, 95% CI 2-sided [-61.58 to -50.68], Standard Error of Mean 2.76
Statistical Analysis 11: Comparison: R40 PBO Q2W vs R40 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -49.17, 95% CI 2-sided [-55.80 to -42.53], Standard Error of Mean 3.36
Statistical Analysis 12: Comparison: R40 PBO QM vs R40 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -48.81, 95% CI 2-sided [-57.21 to -40.40], Standard Error of Mean 4.25
Statistical Analysis 13: Comparison: S40 PBO Q2W vs S40 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -57.73, 95% CI 2-sided [-62.82 to -52.65], Standard Error of Mean 2.57
Statistical Analysis 14: Comparison: S40 PBO QM vs S40 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -52.04, 95% CI 2-sided [-58.10 to -45.98], Standard Error of Mean 3.07

13. Secondary Outcome: Percentage of Participants Who Achieved a Mean LDL-C at Weeks 10 and 12 of Less Than 70 mg/dL
Time Frame: Weeks 10 and 12
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | A10 PBO Q2W | A10 PBO QM | A10 EZE (Q2W) | A10 EZE (QM) | A10 EvoMab Q2W | A10 EvoMab QM | A80 PBO Q2W | A80 PBO QM | A80 EZE (Q2W) | A80 EZE (QM) | A80 EvoMab Q2W | A80 EvoMab QM | R5 PBO Q2W | R5 PBO QM | R5 EvoMab Q2W | R5 EvoMab QM | R40 PBO Q2W | R40 PBO QM | R40 EvoMab Q2W | R40 EvoMab QM | S40 PBO Q2W | S40 PBO QM | S40 EvoMab Q2W | S40 EvoMab QM
Number analyzed (Participants) | 56 | 55 | 56 | 55 | 110 | 110 | 55 | 55 | 56 | 54 | 109 | 110 | 58 | 57 | 113 | 115 | 56 | 55 | 111 | 112 | 56 | 55 | 112 | 115
percentage of participants | 5.7 [1.9 to 15.4] | 5.6 [1.9 to 15.1] | 20.0 [11.2 to 33.0] | 16.7 [9.0 to 28.7] | 88.1 [80.7 to 92.9] | 85.8 [78.0 to 91.2] | 13.7 [6.8 to 25.7] | 9.3 [4.0 to 19.9] | 50.9 [38.1 to 63.6] | 62.3 [48.8 to 74.1] | 94.4 [88.4 to 97.4] | 92.5 [85.9 to 96.2] | 7.0 [2.8 to 16.7] | 5.3 [1.8 to 14.4] | 88.7 [81.2 to 93.4] | 89.9 [82.8 to 94.3] | 38.9 [27.0 to 52.2] | 28.8 [18.3 to 42.3] | 93.5 [87.1 to 96.8] | 94.5 [88.6 to 97.5] | 1.9 [0.3 to 9.8] | 3.9 [1.1 to 13.2] | 93.6 [87.3 to 96.9] | 88.5 [81.3 to 93.2]
Statistical Analysis 1: Comparison: A10 PBO Q2W vs A10 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; Based on Cochran-Mantel Haenszel test stratified by the stratification factors (entry statin therapy and simvastatin contraindicated therapy usage); Treatment Difference = 82.4, 95% CI 2-sided [70.2 to 88.5]
Statistical Analysis 2: Comparison: A10 PBO QM vs A10 EvoMab QM; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 13, analysis 1]; Treatment Difference = 80.3, 95% CI 2-sided [67.9 to 86.8]
Statistical Analysis 3: Comparison: A10 EZE (Q2W) vs A10 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 13, analysis 1]; Treatment Difference = 68.1, 95% CI 2-sided [53.1 to 78.1]
Statistical Analysis 4: Comparison: A10 EZE (QM) vs A10 EvoMab QM; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 13, analysis 1]; Treatment Difference = 69.2, 95% CI 2-sided [54.8 to 78.5]
Statistical Analysis 5: Comparison: A80 PBO Q2W vs A80 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 13, analysis 1]; Treatment Difference = 80.7, 95% CI 2-sided [67.3 to 88.3]
Statistical Analysis 6: Comparison: A80 PBO QM vs A80 EvoMab QM; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 13, analysis 1]; Treatment Difference = 83.3, 95% CI 2-sided [70.7 to 89.6]
Statistical Analysis 7: Comparison: A80 EZE (Q2W) vs A80 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 13, analysis 1]; Treatment Difference = 43.5, 95% CI 2-sided [29.5 to 56.7]
Statistical Analysis 8: Comparison: A80 EZE (QM) vs A80 EvoMab QM; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 13, analysis 1]; Treatment Difference = 30.3, 95% CI 2-sided [16.7 to 44.2]
Statistical Analysis 9: Comparison: R5 PBO Q2W vs R5 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 13, analysis 1]; Treatment Difference = 81.7, 95% CI 2-sided [69.5 to 88.0]
Statistical Analysis 10: Comparison: R5 PBO QM vs R5 EvoMab QM; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 13, analysis 1]; Treatment Difference = 84.6, 95% CI 2-sided [73.1 to 90.2]
Statistical Analysis 11: Comparison: R40 PBO Q2W vs R40 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 13, analysis 1]; Treatment Difference = 54.6, 95% CI 2-sided [39.8 to 66.9]
Statistical Analysis 12: Comparison: R40 PBO QM vs R40 EvoMab QM; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 13, analysis 1]; Treatment Difference = 65.7, 95% CI 2-sided [51.0 to 76.6]
Statistical Analysis 13: Comparison: S40 PBO Q2W vs S40 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 13, analysis 1]; Treatment Difference = 91.7, 95% CI 2-sided [81.6 to 95.3]
Statistical Analysis 14: Comparison: S40 PBO QM vs S40 EvoMab QM; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 13, analysis 1]; Treatment Difference = 84.6, 95% CI 2-sided [72.8 to 90.0]

14. Secondary Outcome: Percentage of Participants Who Achieved LDL-C < 70 mg/dL at Week 12
Time Frame: Week 12
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | A10 PBO Q2W | A10 PBO QM | A10 EZE (Q2W) | A10 EZE (QM) | A10 EvoMab Q2W | A10 EvoMab QM | A80 PBO Q2W | A80 PBO QM | A80 EZE (Q2W) | A80 EZE (QM) | A80 EvoMab Q2W | A80 EvoMab QM | R5 PBO Q2W | R5 PBO QM | R5 EvoMab Q2W | R5 EvoMab QM | R40 PBO Q2W | R40 PBO QM | R40 EvoMab Q2W | R40 EvoMab QM | S40 PBO Q2W | S40 PBO QM | S40 EvoMab Q2W | S40 EvoMab QM
Number analyzed (Participants) | 56 | 55 | 56 | 55 | 110 | 110 | 55 | 55 | 56 | 54 | 109 | 110 | 58 | 57 | 113 | 115 | 56 | 55 | 111 | 112 | 56 | 55 | 112 | 115
percentage of participants | 2.0 [0.3 to 10.3] | 5.9 [2.0 to 15.9] | 22.4 [13.0 to 35.9] | 19.2 [10.8 to 31.9] | 85.4 [77.4 to 91.0] | 84.2 [75.8 to 90.0] | 13.0 [6.1 to 25.7] | 9.8 [4.3 to 21.0] | 52.0 [38.5 to 65.2] | 55.8 [42.3 to 68.4] | 93.1 [86.5 to 96.6] | 91.0 [83.8 to 95.2] | 7.7 [3.0 to 18.2] | 5.5 [1.9 to 14.9] | 85.0 [76.7 to 90.7] | 86.5 [78.7 to 91.8] | 39.6 [27.6 to 53.1] | 28.0 [17.5 to 41.7] | 92.3 [85.6 to 96.1] | 92.3 [85.6 to 96.1] | 1.9 [0.3 to 10.1] | 6.4 [2.2 to 17.2] | 94.4 [88.4 to 97.4] | 84.8 [76.7 to 90.4]
Statistical Analysis 1: Comparison: A10 PBO Q2W vs A10 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 13, analysis 1]; Treatment Difference = 83.5, 95% CI 2-sided [71.9 to 89.2]
Statistical Analysis 2: Comparison: A10 PBO QM vs A10 EvoMab QM; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 13, analysis 1]; Treatment Difference = 78.3, 95% CI 2-sided [65.2 to 85.3]
Statistical Analysis 3: Comparison: A10 EZE (Q2W) vs A10 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 13, analysis 1]; Treatment Difference = 63.0, 95% CI 2-sided [47.3 to 73.9]
Statistical Analysis 4: Comparison: A10 EZE (QM) vs A10 EvoMab QM; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 13, analysis 1]; Treatment Difference = 64.9, 95% CI 2-sided [49.8 to 75.2]
Statistical Analysis 5: Comparison: A80 PBO Q2W vs A80 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 13, analysis 1]; Treatment Difference = 80.1, 95% CI 2-sided [65.8 to 87.9]
Statistical Analysis 6: Comparison: A80 PBO QM vs A80 EvoMab QM; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 13, analysis 1]; Treatment Difference = 81.2, 95% CI 2-sided [67.9 to 88.1]
Statistical Analysis 7: Comparison: A80 EZE (Q2W) vs A80 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 13, analysis 1]; Treatment Difference = 41.1, 95% CI 2-sided [26.4 to 55.1]
Statistical Analysis 8: Comparison: A80 EZE (QM) vs A80 EvoMab QM; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 13, analysis 1]; Treatment Difference = 35.2, 95% CI 2-sided [20.7 to 49.3]
Statistical Analysis 9: Comparison: R5 PBO Q2W vs R5 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 13, analysis 1]; Treatment Difference = 77.3, 95% CI 2-sided [63.9 to 84.7]
Statistical Analysis 10: Comparison: R5 PBO QM vs R5 EvoMab QM; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 13, analysis 1]; Treatment Difference = 81.1, 95% CI 2-sided [68.8 to 87.5]
Statistical Analysis 11: Comparison: R40 PBO Q2W vs R40 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 13, analysis 1]; Treatment Difference = 52.7, 95% CI 2-sided [37.6 to 65.3]
Statistical Analysis 12: Comparison: R40 PBO QM vs R40 EvoMab QM; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 13, analysis 1]; Treatment Difference = 64.3, 95% CI 2-sided [49.1 to 75.5]
Statistical Analysis 13: Comparison: S40 PBO Q2W vs S40 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 13, analysis 1]; Treatment Difference = 92.5, 95% CI 2-sided [82.3 to 95.9]
Statistical Analysis 14: Comparison: S40 PBO QM vs S40 EvoMab QM; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 13, analysis 1]; Treatment Difference = 78.4, 95% CI 2-sided [64.9 to 85.4]

15. Secondary Outcome: Percent Change From Baseline in Lipoprotein(a) at the Mean of Weeks 10 and 12
Time Frame: Baseline and Weeks 10 and 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | A10 PBO Q2W | A10 PBO QM | A10 EZE (Q2W) | A10 EZE (QM) | A10 EvoMab Q2W | A10 EvoMab QM | A80 PBO Q2W | A80 PBO QM | A80 EZE (Q2W) | A80 EZE (QM) | A80 EvoMab Q2W | A80 EvoMab QM | R5 PBO Q2W | R5 PBO QM | R5 EvoMab Q2W | R5 EvoMab QM | R40 PBO Q2W | R40 PBO QM | R40 EvoMab Q2W | R40 EvoMab QM | S40 PBO Q2W | S40 PBO QM | S40 EvoMab Q2W | S40 EvoMab QM
Number analyzed (Participants) | 56 | 55 | 56 | 55 | 110 | 110 | 55 | 55 | 56 | 54 | 109 | 110 | 58 | 57 | 113 | 115 | 56 | 55 | 111 | 112 | 56 | 55 | 112 | 115
percent change | 6.07 (2.86) | -0.77 (3.28) | 1.44 (3.02) | 6.85 (3.29) | -26.01 (2.08) | -22.64 (2.27) | -3.45 (2.99) | 1.51 (3.35) | 8.05 (2.94) | 9.96 (3.40) | -23.97 (2.10) | -27.46 (2.39) | 11.41 (3.00) | 3.65 (3.56) | -24.26 (2.21) | -23.16 (2.50) | 8.59 (2.98) | 6.26 (3.59) | -24.96 (2.12) | -25.93 (2.46) | -10.57 (4.49) | -4.99 (5.37) | -38.64 (3.92) | -32.16 (4.50)
Statistical Analysis 1: Comparison: A10 PBO Q2W vs A10 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -32.08, 95% CI 2-sided [-39.06 to -25.11], Standard Error of Mean 3.54
Statistical Analysis 2: Comparison: A10 PBO QM vs A10 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -21.86, 95% CI 2-sided [-29.70 to -14.03], Standard Error of Mean 3.98
Statistical Analysis 3: Comparison: A10 EZE (Q2W) vs A10 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -27.45, 95% CI 2-sided [-34.53 to -20.38], Standard Error of Mean 3.59
Statistical Analysis 4: Comparison: A10 EZE (QM) vs A10 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -29.49, 95% CI 2-sided [-37.36 to -21.62], Standard Error of Mean 3.99
Statistical Analysis 5: Comparison: A80 PBO Q2W vs A80 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -20.52, 95% CI 2-sided [-27.71 to -13.33], Standard Error of Mean 3.65
Statistical Analysis 6: Comparison: A80 PBO QM vs A80 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -28.96, 95% CI 2-sided [-37.01 to -20.92], Standard Error of Mean 4.08
Statistical Analysis 7: Comparison: A80 EZE (Q2W) vs A80 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -32.02, 95% CI 2-sided [-39.11 to -24.93], Standard Error of Mean 3.60
Statistical Analysis 8: Comparison: A80 EZE (QM) vs A80 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -37.42, 95% CI 2-sided [-45.61 to -29.23], Standard Error of Mean 4.15
Statistical Analysis 9: Comparison: R5 PBO Q2W vs R5 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -35.66, 95% CI 2-sided [-42.94 to -28.38], Standard Error of Mean 3.69
Statistical Analysis 10: Comparison: R5 PBO QM vs R5 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -26.81, 95% CI 2-sided [-35.36 to -18.27], Standard Error of Mean 4.33
Statistical Analysis 11: Comparison: R40 PBO Q2W vs R40 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -33.56, 95% CI 2-sided [-40.74 to -26.37], Standard Error of Mean 3.64
Statistical Analysis 12: Comparison: R40 PBO QM vs R40 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -32.19, 95% CI 2-sided [-40.80 to -23.58], Standard Error of Mean 4.36
Statistical Analysis 13: Comparison: S40 PBO Q2W vs S40 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -28.07, 95% CI 2-sided [-34.91 to -21.23], Standard Error of Mean 3.46
Statistical Analysis 14: Comparison: S40 PBO QM vs S40 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -27.16, 95% CI 2-sided [-34.59 to -19.73], Standard Error of Mean 3.76

16. Secondary Outcome: Percent Change From Baseline in Lipoprotein(a) at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | A10 PBO Q2W | A10 PBO QM | A10 EZE (Q2W) | A10 EZE (QM) | A10 EvoMab Q2W | A10 EvoMab QM | A80 PBO Q2W | A80 PBO QM | A80 EZE (Q2W) | A80 EZE (QM) | A80 EvoMab Q2W | A80 EvoMab QM | R5 PBO Q2W | R5 PBO QM | R5 EvoMab Q2W | R5 EvoMab QM | R40 PBO Q2W | R40 PBO QM | R40 EvoMab Q2W | R40 EvoMab QM | S40 PBO Q2W | S40 PBO QM | S40 EvoMab Q2W | S40 EvoMab QM
Number analyzed (Participants) | 56 | 55 | 56 | 55 | 110 | 110 | 55 | 55 | 56 | 54 | 109 | 110 | 58 | 57 | 113 | 115 | 56 | 55 | 111 | 112 | 56 | 55 | 112 | 115
percent change | 7.34 (3.13) | -0.43 (3.38) | 3.29 (3.28) | 7.18 (3.38) | -25.87 (2.26) | -20.25 (2.36) | -2.23 (3.35) | 3.41 (3.54) | 8.01 (3.26) | 10.20 (3.57) | -24.61 (2.31) | -24.68 (2.53) | 11.40 (3.37) | 4.49 (3.68) | -25.09 (2.47) | -20.85 (2.59) | 10.38 (3.09) | 10.21 (4.36) | -26.11 (2.21) | -21.97 (2.97) | -6.81 (4.57) | -1.06 (5.67) | -38.06 (3.96) | -29.23 (4.68)
Statistical Analysis 1: Comparison: A10 PBO Q2W vs A10 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -33.20, 95% CI 2-sided [-40.81 to -25.60], Standard Error of Mean 3.86
Statistical Analysis 2: Comparison: A10 PBO QM vs A10 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -19.82, 95% CI 2-sided [-27.92 to -11.72], Standard Error of Mean 4.11
Statistical Analysis 3: Comparison: A10 EZE (Q2W) vs A10 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -29.16, 95% CI 2-sided [-36.87 to -21.44], Standard Error of Mean 3.91
Statistical Analysis 4: Comparison: A10 EZE (QM) vs A10 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -27.44, 95% CI 2-sided [-35.56 to -19.32], Standard Error of Mean 4.12
Statistical Analysis 5: Comparison: A80 PBO Q2W vs A80 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -22.38, 95% CI 2-sided [-30.39 to -14.36], Standard Error of Mean 4.07
Statistical Analysis 6: Comparison: A80 PBO QM vs A80 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -28.10, 95% CI 2-sided [-36.62 to -19.58], Standard Error of Mean 4.32
Statistical Analysis 7: Comparison: A80 EZE (Q2W) vs A80 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -32.62, 95% CI 2-sided [-40.46 to -24.78], Standard Error of Mean 3.98
Statistical Analysis 8: Comparison: A80 EZE (QM) vs A80 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -34.88, 95% CI 2-sided [-43.52 to -26.25], Standard Error of Mean 4.38
Statistical Analysis 9: Comparison: R5 PBO Q2W vs R5 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -36.50, 95% CI 2-sided [-44.69 to -28.30], Standard Error of Mean 4.15
Statistical Analysis 10: Comparison: R5 PBO QM vs R5 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -25.34, 95% CI 2-sided [-34.19 to -16.49], Standard Error of Mean 4.48
Statistical Analysis 11: Comparison: R40 PBO Q2W vs R40 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -36.48, 95% CI 2-sided [-43.95 to -29.02], Standard Error of Mean 3.78
Statistical Analysis 12: Comparison: R40 PBO QM vs R40 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -32.17, 95% CI 2-sided [-42.61 to -21.74], Standard Error of Mean 5.28
Statistical Analysis 13: Comparison: S40 PBO Q2W vs S40 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -31.25, 95% CI 2-sided [-38.40 to -24.10], Standard Error of Mean 3.62
Statistical Analysis 14: Comparison: S40 PBO QM vs S40 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -28.17, 95% CI 2-sided [-36.79 to -19.55], Standard Error of Mean 4.36

17. Secondary Outcome: Percent Change From Baseline in Triglycerides at the Mean of Weeks 10 and 12
Time Frame: Baseline and Weeks 10 and 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | A10 PBO Q2W | A10 PBO QM | A10 EZE (Q2W) | A10 EZE (QM) | A10 EvoMab Q2W | A10 EvoMab QM | A80 PBO Q2W | A80 PBO QM | A80 EZE (Q2W) | A80 EZE (QM) | A80 EvoMab Q2W | A80 EvoMab QM | R5 PBO Q2W | R5 PBO QM | R5 EvoMab Q2W | R5 EvoMab QM | R40 PBO Q2W | R40 PBO QM | R40 EvoMab Q2W | R40 EvoMab QM | S40 PBO Q2W | S40 PBO QM | S40 EvoMab Q2W | S40 EvoMab QM
Number analyzed (Participants) | 56 | 55 | 56 | 55 | 110 | 110 | 55 | 55 | 56 | 54 | 109 | 110 | 58 | 57 | 113 | 115 | 56 | 55 | 111 | 112 | 56 | 55 | 112 | 115
percent change | 6.49 (3.94) | 9.17 (4.41) | -3.16 (4.10) | 1.57 (4.35) | -5.61 (2.81) | -13.38 (3.08) | 6.16 (4.02) | 8.05 (4.35) | -8.10 (3.92) | -4.86 (4.39) | -9.27 (2.80) | -6.36 (3.11) | 12.43 (4.19) | 12.26 (4.67) | -10.28 (3.04) | -7.26 (3.29) | 8.44 (3.76) | 10.75 (3.98) | -9.15 (2.70) | -15.43 (2.77) | 9.29 (6.97) | 13.78 (7.44) | -11.67 (5.97) | -15.93 (6.15)
Statistical Analysis 1: Comparison: A10 PBO Q2W vs A10 EvoMab Q2W; Test type: Superiority or Other; p = 0.20, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -12.10, 95% CI 2-sided [-21.63 to -2.58], Standard Error of Mean 4.83
Statistical Analysis 2: Comparison: A10 PBO QM vs A10 EvoMab QM; Test type: Superiority or Other; p = 0.003, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -22.55, 95% CI 2-sided [-33.13 to -11.97], Standard Error of Mean 5.36
Statistical Analysis 3: Comparison: A10 EZE (Q2W) vs A10 EvoMab Q2W; Test type: Superiority or Other; p = 1.00, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -2.45, 95% CI 2-sided [-12.09 to 7.19], Standard Error of Mean 4.89
Statistical Analysis 4: Comparison: A10 EZE (QM) vs A10 EvoMab QM; Test type: Superiority or Other; p = 0.053, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -14.95, 95% CI 2-sided [-25.46 to -4.44], Standard Error of Mean 5.33
Statistical Analysis 5: Comparison: A80 PBO Q2W vs A80 EvoMab Q2W; Test type: Superiority or Other; p = 0.073, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -15.43, 95% CI 2-sided [-25.06 to -5.79], Standard Error of Mean 4.89
Statistical Analysis 6: Comparison: A80 PBO QM vs A80 EvoMab QM; Test type: Superiority or Other; p = 0.027, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -14.41, 95% CI 2-sided [-24.90 to -3.92], Standard Error of Mean 5.32
Statistical Analysis 7: Comparison: A80 EZE (Q2W) vs A80 EvoMab Q2W; Test type: Superiority or Other; p = 1.00, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -1.17, 95% CI 2-sided [-10.63 to 8.30], Standard Error of Mean 4.80
Statistical Analysis 8: Comparison: A80 EZE (QM) vs A80 EvoMab QM; Test type: Superiority or Other; p = 0.63, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -1.51, 95% CI 2-sided [-12.12 to 9.11], Standard Error of Mean 5.38
Statistical Analysis 9: Comparison: R5 PBO Q2W vs R5 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -22.72, 95% CI 2-sided [-32.90 to -12.54], Standard Error of Mean 5.15
Statistical Analysis 10: Comparison: R5 PBO QM vs R5 EvoMab QM; Test type: Superiority or Other; p = 0.007, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -19.52, 95% CI 2-sided [-30.76 to -8.28], Standard Error of Mean 5.69
Statistical Analysis 11: Comparison: R40 PBO Q2W vs R40 EvoMab Q2W; Test type: Superiority or Other; p = 0.002, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -17.59, 95% CI 2-sided [-26.71 to -8.46], Standard Error of Mean 4.62
Statistical Analysis 12: Comparison: R40 PBO QM vs R40 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -26.18, 95% CI 2-sided [-35.76 to -16.59], Standard Error of Mean 4.85
Statistical Analysis 13: Comparison: S40 PBO Q2W vs S40 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -20.97, 95% CI 2-sided [-32.38 to -9.55], Standard Error of Mean 5.78
Statistical Analysis 14: Comparison: S40 PBO QM vs S40 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -29.71, 95% CI 2-sided [-40.84 to -18.57], Standard Error of Mean 5.64

18. Secondary Outcome: Percent Change From Baseline in Triglycerides at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | A10 PBO Q2W | A10 PBO QM | A10 EZE (Q2W) | A10 EZE (QM) | A10 EvoMab Q2W | A10 EvoMab QM | A80 PBO Q2W | A80 PBO QM | A80 EZE (Q2W) | A80 EZE (QM) | A80 EvoMab Q2W | A80 EvoMab QM | R5 PBO Q2W | R5 PBO QM | R5 EvoMab Q2W | R5 EvoMab QM | R40 PBO Q2W | R40 PBO QM | R40 EvoMab Q2W | R40 EvoMab QM | S40 PBO Q2W | S40 PBO QM | S40 EvoMab Q2W | S40 EvoMab QM
Number analyzed (Participants) | 56 | 55 | 56 | 55 | 110 | 110 | 55 | 55 | 56 | 54 | 109 | 110 | 58 | 57 | 113 | 115 | 56 | 55 | 111 | 112 | 56 | 55 | 112 | 115
percent change | 8.27 (5.23) | 14.35 (5.92) | -0.43 (5.39) | 4.88 (5.84) | -3.79 (3.72) | -13.26 (4.17) | 6.65 (4.45) | 8.22 (5.22) | -7.40 (4.32) | -3.11 (5.23) | -10.07 (3.05) | -1.10 (3.74) | 13.57 (5.76) | 12.96 (5.32) | -4.46 (4.16) | -6.88 (3.80) | 10.97 (4.66) | 10.00 (4.38) | -5.58 (3.34) | -10.51 (3.04) | 8.07 (6.88) | 16.72 (7.88) | -13.71 (5.91) | -14.65 (6.39)
Statistical Analysis 1: Comparison: A10 PBO Q2W vs A10 EvoMab Q2W; Test type: Superiority or Other; p = 0.20, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -12.06, 95% CI 2-sided [-24.69 to 0.57], Standard Error of Mean 6.41
Statistical Analysis 2: Comparison: A10 PBO QM vs A10 EvoMab QM; Test type: Superiority or Other; p = 0.003, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -27.60, 95% CI 2-sided [-41.86 to -13.35], Standard Error of Mean 7.23
Statistical Analysis 3: Comparison: A10 EZE (Q2W) vs A10 EvoMab Q2W; Test type: Superiority or Other; p = 1.00, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -3.37, 95% CI 2-sided [-16.16 to 9.43], Standard Error of Mean 6.49
Statistical Analysis 4: Comparison: A10 EZE (QM) vs A10 EvoMab QM; Test type: Superiority or Other; p = 0.053, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -18.13, 95% CI 2-sided [-32.28 to -3.99], Standard Error of Mean 7.18
Statistical Analysis 5: Comparison: A80 PBO Q2W vs A80 EvoMab Q2W; Test type: Superiority or Other; p = 0.073, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -16.72, 95% CI 2-sided [-27.34 to -6.10], Standard Error of Mean 5.39
Statistical Analysis 6: Comparison: A80 PBO QM vs A80 EvoMab QM; Test type: Superiority or Other; p = 0.027, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -9.31, 95% CI 2-sided [-21.92 to 3.29], Standard Error of Mean 6.39
Statistical Analysis 7: Comparison: A80 EZE (Q2W) vs A80 EvoMab Q2W; Test type: Superiority or Other; p = 1.00, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -2.67, 95% CI 2-sided [-13.05 to 7.72], Standard Error of Mean 5.27
Statistical Analysis 8: Comparison: A80 EZE (QM) vs A80 EvoMab QM; Test type: Superiority or Other; p = 0.63, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 2.02, 95% CI 2-sided [-10.66 to 14.69], Standard Error of Mean 6.43
Statistical Analysis 9: Comparison: R5 PBO Q2W vs R5 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -18.03, 95% CI 2-sided [-32.03 to -4.04], Standard Error of Mean 7.08
Statistical Analysis 10: Comparison: R5 PBO QM vs R5 EvoMab QM; Test type: Superiority or Other; p = 0.007, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -19.83, 95% CI 2-sided [-32.71 to -6.96], Standard Error of Mean 6.52
Statistical Analysis 11: Comparison: R40 PBO Q2W vs R40 EvoMab Q2W; Test type: Superiority or Other; p = 0.002, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -16.55, 95% CI 2-sided [-27.84 to -5.26], Standard Error of Mean 5.71
Statistical Analysis 12: Comparison: R40 PBO QM vs R40 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -20.51, 95% CI 2-sided [-31.04 to -9.98], Standard Error of Mean 5.33
Statistical Analysis 13: Comparison: S40 PBO Q2W vs S40 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -21.78, 95% CI 2-sided [-32.88 to -10.68], Standard Error of Mean 5.62
Statistical Analysis 14: Comparison: S40 PBO QM vs S40 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -31.36, 95% CI 2-sided [-44.10 to -18.62], Standard Error of Mean 6.45

19. Secondary Outcome: Percent Change From Baseline in Very Low-Density Cholesterol (VLDL-C) at the Mean of Weeks 10 and 12
Time Frame: Baseline and Weeks 10 and 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | A10 PBO Q2W | A10 PBO QM | A10 EZE (Q2W) | A10 EZE (QM) | A10 EvoMab Q2W | A10 EvoMab QM | A80 PBO Q2W | A80 PBO QM | A80 EZE (Q2W) | A80 EZE (QM) | A80 EvoMab Q2W | A80 EvoMab QM | R5 PBO Q2W | R5 PBO QM | R5 EvoMab Q2W | R5 EvoMab QM | R40 PBO Q2W | R40 PBO QM | R40 EvoMab Q2W | R40 EvoMab QM | S40 PBO Q2W | S40 PBO QM | S40 EvoMab Q2W | S40 EvoMab QM
Number analyzed (Participants) | 56 | 55 | 56 | 55 | 110 | 110 | 55 | 55 | 56 | 54 | 109 | 110 | 58 | 57 | 113 | 115 | 56 | 55 | 111 | 112 | 56 | 55 | 112 | 115
percent change | 6.51 (3.56) | 9.53 (4.45) | -5.35 (3.74) | 1.77 (4.41) | -6.85 (2.56) | -11.77 (3.11) | 6.24 (4.03) | 8.31 (4.26) | -8.52 (3.93) | -6.13 (4.31) | -8.96 (2.82) | -6.38 (3.05) | 12.86 (3.95) | 12.54 (4.58) | -12.22 (2.86) | -7.25 (3.23) | 7.06 (3.76) | 8.13 (3.72) | -9.09 (2.71) | -15.05 (2.58) | 8.64 (6.01) | 16.37 (7.15) | -14.57 (5.17) | -16.50 (5.87)
Statistical Analysis 1: Comparison: A10 PBO Q2W vs A10 EvoMab Q2W; Test type: Superiority or Other; p = 0.088, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -13.36, 95% CI 2-sided [-21.99 to -4.74], Standard Error of Mean 4.38
Statistical Analysis 2: Comparison: A10 PBO QM vs A10 EvoMab QM; Test type: Superiority or Other; p = 0.005, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -21.31, 95% CI 2-sided [-31.98 to -10.64], Standard Error of Mean 5.41
Statistical Analysis 3: Comparison: A10 EZE (Q2W) vs A10 EvoMab Q2W; Test type: Superiority or Other; p = 1.00, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -1.50, 95% CI 2-sided [-10.27 to 7.27], Standard Error of Mean 4.45
Statistical Analysis 4: Comparison: A10 EZE (QM) vs A10 EvoMab QM; Test type: Superiority or Other; p = 0.056, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -13.54, 95% CI 2-sided [-24.17 to -2.91], Standard Error of Mean 5.39
Statistical Analysis 5: Comparison: A80 PBO Q2W vs A80 EvoMab Q2W; Test type: Superiority or Other; p = 0.073, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -15.21, 95% CI 2-sided [-24.88 to -5.54], Standard Error of Mean 4.91
Statistical Analysis 6: Comparison: A80 PBO QM vs A80 EvoMab QM; Test type: Superiority or Other; p = 0.027, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -14.69, 95% CI 2-sided [-24.97 to -4.42], Standard Error of Mean 5.21
Statistical Analysis 7: Comparison: A80 EZE (Q2W) vs A80 EvoMab Q2W; Test type: Superiority or Other; p = 1.00, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -0.44, 95% CI 2-sided [-9.94 to 9.05], Standard Error of Mean 4.82
Statistical Analysis 8: Comparison: A80 EZE (QM) vs A80 EvoMab QM; Test type: Superiority or Other; p = 0.62, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -0.25, 95% CI 2-sided [-10.66 to 10.16], Standard Error of Mean 5.28
Statistical Analysis 9: Comparison: R5 PBO Q2W vs R5 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -25.07, 95% CI 2-sided [-34.64 to -15.50], Standard Error of Mean 4.85
Statistical Analysis 10: Comparison: R5 PBO QM vs R5 EvoMab QM; Test type: Superiority or Other; p = 0.007, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -19.79, 95% CI 2-sided [-30.81 to -8.77], Standard Error of Mean 5.58
Statistical Analysis 11: Comparison: R40 PBO Q2W vs R40 EvoMab Q2W; Test type: Superiority or Other; p = 0.005, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -16.15, 95% CI 2-sided [-25.27 to -7.03], Standard Error of Mean 4.61
Statistical Analysis 12: Comparison: R40 PBO QM vs R40 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -23.18, 95% CI 2-sided [-32.11 to -14.25], Standard Error of Mean 4.52
Statistical Analysis 13: Comparison: S40 PBO Q2W vs S40 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -23.21, 95% CI 2-sided [-33.00 to -13.43], Standard Error of Mean 4.95
Statistical Analysis 14: Comparison: S40 PBO QM vs S40 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -32.87, 95% CI 2-sided [-43.60 to -22.14], Standard Error of Mean 5.43

20. Secondary Outcome: Percent Change From Baseline in Very Low-Density Cholesterol (VLDL-C) at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | A10 PBO Q2W | A10 PBO QM | A10 EZE (Q2W) | A10 EZE (QM) | A10 EvoMab Q2W | A10 EvoMab QM | A80 PBO Q2W | A80 PBO QM | A80 EZE (Q2W) | A80 EZE (QM) | A80 EvoMab Q2W | A80 EvoMab QM | R5 PBO Q2W | R5 PBO QM | R5 EvoMab Q2W | R5 EvoMab QM | R40 PBO Q2W | R40 PBO QM | R40 EvoMab Q2W | R40 EvoMab QM | S40 PBO Q2W | S40 PBO QM | S40 EvoMab Q2W | S40 EvoMab QM
Number analyzed (Participants) | 56 | 55 | 56 | 55 | 110 | 110 | 55 | 55 | 56 | 54 | 109 | 110 | 58 | 57 | 113 | 115 | 56 | 55 | 111 | 112 | 56 | 55 | 112 | 115
percent change | 8.32 (4.00) | 14.74 (5.91) | -4.61 (4.19) | 3.45 (5.89) | -6.16 (2.88) | -11.73 (4.16) | 6.73 (4.45) | 8.54 (5.00) | -7.92 (4.32) | -6.00 (5.04) | -9.69 (3.05) | -1.06 (3.58) | 13.79 (5.05) | 12.47 (5.31) | -8.20 (3.64) | -6.28 (3.78) | 10.09 (4.65) | 8.59 (4.37) | -6.10 (3.33) | -9.95 (3.03) | 7.63 (6.26) | 20.97 (7.53) | -14.83 (5.30) | -15.86 (6.09)
Statistical Analysis 1: Comparison: A10 PBO Q2W vs A10 EvoMab Q2W; Test type: Superiority or Other; p = 0.088, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -14.47, 95% CI 2-sided [-24.16 to -4.78], Standard Error of Mean 4.92
Statistical Analysis 2: Comparison: A10 PBO QM vs A10 EvoMab QM; Test type: Superiority or Other; p = 0.005, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -26.47, 95% CI 2-sided [-40.71 to -12.24], Standard Error of Mean 7.22
Statistical Analysis 3: Comparison: A10 EZE (Q2W) vs A10 EvoMab Q2W; Test type: Superiority or Other; p = 1.00, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -1.54, 95% CI 2-sided [-11.41 to 8.32], Standard Error of Mean 5.00
Statistical Analysis 4: Comparison: A10 EZE (QM) vs A10 EvoMab QM; Test type: Superiority or Other; p = 0.056, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -15.19, 95% CI 2-sided [-29.40 to -0.97], Standard Error of Mean 7.21
Statistical Analysis 5: Comparison: A80 PBO Q2W vs A80 EvoMab Q2W; Test type: Superiority or Other; p = 0.073, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -16.42, 95% CI 2-sided [-27.05 to -5.80], Standard Error of Mean 5.39
Statistical Analysis 6: Comparison: A80 PBO QM vs A80 EvoMab QM; Test type: Superiority or Other; p = 0.027, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -9.60, 95% CI 2-sided [-21.68 to 2.48], Standard Error of Mean 6.13
Statistical Analysis 7: Comparison: A80 EZE (Q2W) vs A80 EvoMab Q2W; Test type: Superiority or Other; p = 1.00, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -1.78, 95% CI 2-sided [-12.16 to 8.61], Standard Error of Mean 5.27
Statistical Analysis 8: Comparison: A80 EZE (QM) vs A80 EvoMab QM; Test type: Superiority or Other; p = 0.62, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 4.94, 95% CI 2-sided [-7.25 to 17.14], Standard Error of Mean 6.18
Statistical Analysis 9: Comparison: R5 PBO Q2W vs R5 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -21.98, 95% CI 2-sided [-34.24 to -9.73], Standard Error of Mean 6.20
Statistical Analysis 10: Comparison: R5 PBO QM vs R5 EvoMab QM; Test type: Superiority or Other; p = 0.007, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -18.75, 95% CI 2-sided [-31.60 to -5.90], Standard Error of Mean 6.50
Statistical Analysis 11: Comparison: R40 PBO Q2W vs R40 EvoMab Q2W; Test type: Superiority or Other; p = 0.005, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -16.19, 95% CI 2-sided [-27.46 to -4.92], Standard Error of Mean 5.70
Statistical Analysis 12: Comparison: R40 PBO QM vs R40 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -18.54, 95% CI 2-sided [-29.04 to -8.05], Standard Error of Mean 5.31
Statistical Analysis 13: Comparison: S40 PBO Q2W vs S40 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -22.45, 95% CI 2-sided [-33.09 to -11.81], Standard Error of Mean 5.39
Statistical Analysis 14: Comparison: S40 PBO QM vs S40 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -36.83, 95% CI 2-sided [-48.96 to -24.70], Standard Error of Mean 6.14

21. Secondary Outcome: Percent Change From Baseline in HDL-C at the Mean of Weeks 10 and 12
Time Frame: Baseline and Weeks 10 and 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | A10 PBO Q2W | A10 PBO QM | A10 EZE (Q2W) | A10 EZE (QM) | A10 EvoMab Q2W | A10 EvoMab QM | A80 PBO Q2W | A80 PBO QM | A80 EZE (Q2W) | A80 EZE (QM) | A80 EvoMab Q2W | A80 EvoMab QM | R5 PBO Q2W | R5 PBO QM | R5 EvoMab Q2W | R5 EvoMab QM | R40 PBO Q2W | R40 PBO QM | R40 EvoMab Q2W | R40 EvoMab QM | S40 PBO Q2W | S40 PBO QM | S40 EvoMab Q2W | S40 EvoMab QM
Number analyzed (Participants) | 56 | 55 | 56 | 55 | 110 | 110 | 55 | 55 | 56 | 54 | 109 | 110 | 58 | 57 | 113 | 115 | 56 | 55 | 111 | 112 | 56 | 55 | 112 | 115
percent change | -0.99 (1.50) | -0.45 (1.94) | -1.13 (1.56) | -0.92 (1.92) | 5.54 (1.07) | 7.66 (1.37) | 4.48 (1.73) | -1.37 (1.85) | 0.86 (1.68) | -0.59 (1.86) | 8.44 (1.20) | 7.76 (1.31) | 0.87 (1.52) | -0.94 (2.55) | 6.23 (1.10) | 7.72 (1.80) | -0.60 (1.56) | -0.40 (1.81) | 4.86 (1.12) | 6.35 (1.26) | 0.13 (2.75) | -2.14 (2.72) | 10.35 (2.26) | 6.71 (2.25)
Statistical Analysis 1: Comparison: A10 PBO Q2W vs A10 EvoMab Q2W; Test type: Superiority or Other; p = 0.034, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 6.53, 95% CI 2-sided [2.91 to 10.15], Standard Error of Mean 1.84
Statistical Analysis 2: Comparison: A10 PBO QM vs A10 EvoMab QM; Test type: Superiority or Other; p = 0.017, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 8.11, 95% CI 2-sided [3.43 to 12.79], Standard Error of Mean 2.37
Statistical Analysis 3: Comparison: A10 EZE (Q2W) vs A10 EvoMab Q2W; Test type: Superiority or Other; p = 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 6.67, 95% CI 2-sided [3.00 to 10.34], Standard Error of Mean 1.86
Statistical Analysis 4: Comparison: A10 EZE (QM) vs A10 EvoMab QM; Test type: Superiority or Other; p = 0.006, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 8.57, 95% CI 2-sided [3.93 to 13.22], Standard Error of Mean 2.36
Statistical Analysis 5: Comparison: A80 PBO Q2W vs A80 EvoMab Q2W; Test type: Superiority or Other; p = 0.85, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 3.95, 95% CI 2-sided [-0.19 to 8.09], Standard Error of Mean 2.10
Statistical Analysis 6: Comparison: A80 PBO QM vs A80 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 9.13, 95% CI 2-sided [4.68 to 13.58], Standard Error of Mean 2.26
Statistical Analysis 7: Comparison: A80 EZE (Q2W) vs A80 EvoMab Q2W; Test type: Superiority or Other; p = 0.003, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 7.57, 95% CI 2-sided [3.51 to 11.64], Standard Error of Mean 2.06
Statistical Analysis 8: Comparison: A80 EZE (QM) vs A80 EvoMab QM; Test type: Superiority or Other; p = 0.003, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 8.35, 95% CI 2-sided [3.86 to 12.84], Standard Error of Mean 2.28
Statistical Analysis 9: Comparison: R5 PBO Q2W vs R5 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 5.36, 95% CI 2-sided [1.68 to 9.04], Standard Error of Mean 1.87
Statistical Analysis 10: Comparison: R5 PBO QM vs R5 EvoMab QM; Test type: Superiority or Other; p = 0.010, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 8.66, 95% CI 2-sided [2.51 to 14.80], Standard Error of Mean 3.11
Statistical Analysis 11: Comparison: R40 PBO Q2W vs R40 EvoMab Q2W; Test type: Superiority or Other; p = 0.013, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 5.46, 95% CI 2-sided [1.69 to 9.23], Standard Error of Mean 1.91
Statistical Analysis 12: Comparison: R40 PBO QM vs R40 EvoMab QM; Test type: Superiority or Other; p = 0.002, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 6.75, 95% CI 2-sided [2.40 to 11.10], Standard Error of Mean 2.20
Statistical Analysis 13: Comparison: S40 PBO Q2W vs S40 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 10.23, 95% CI 2-sided [5.13 to 15.32], Standard Error of Mean 2.58
Statistical Analysis 14: Comparison: S40 PBO QM vs S40 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 8.85, 95% CI 2-sided [4.73 to 12.97], Standard Error of Mean 2.09

22. Secondary Outcome: Percent Change From Baseline in HDL-C at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | A10 PBO Q2W | A10 PBO QM | A10 EZE (Q2W) | A10 EZE (QM) | A10 EvoMab Q2W | A10 EvoMab QM | A80 PBO Q2W | A80 PBO QM | A80 EZE (Q2W) | A80 EZE (QM) | A80 EvoMab Q2W | A80 EvoMab QM | R5 PBO Q2W | R5 PBO QM | R5 EvoMab Q2W | R5 EvoMab QM | R40 PBO Q2W | R40 PBO QM | R40 EvoMab Q2W | R40 EvoMab QM | S40 PBO Q2W | S40 PBO QM | S40 EvoMab Q2W | S40 EvoMab QM
Number analyzed (Participants) | 56 | 55 | 56 | 55 | 110 | 110 | 55 | 55 | 56 | 54 | 109 | 110 | 58 | 57 | 113 | 115 | 56 | 55 | 111 | 112 | 56 | 55 | 112 | 115
percent change | 0.22 (1.72) | 0.01 (2.02) | -1.76 (1.78) | -0.40 (1.99) | 7.04 (1.23) | 7.88 (1.42) | 5.02 (1.88) | 0.30 (2.01) | 0.62 (1.83) | 0.21 (2.01) | 9.09 (1.29) | 7.36 (1.43) | 2.87 (1.87) | -0.16 (2.64) | 6.07 (1.35) | 7.18 (1.87) | -0.39 (1.86) | 0.73 (1.98) | 4.65 (1.34) | 5.57 (1.37) | 1.14 (2.96) | -2.65 (2.87) | 10.92 (2.38) | 6.41 (2.34)
Statistical Analysis 1: Comparison: A10 PBO Q2W vs A10 EvoMab Q2W; Test type: Superiority or Other; p = 0.034, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 6.83, 95% CI 2-sided [2.66 to 10.99], Standard Error of Mean 2.11
Statistical Analysis 2: Comparison: A10 PBO QM vs A10 EvoMab QM; Test type: Superiority or Other; p = 0.017, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 7.87, 95% CI 2-sided [3.01 to 12.73], Standard Error of Mean 2.46
Statistical Analysis 3: Comparison: A10 EZE (Q2W) vs A10 EvoMab Q2W; Test type: Superiority or Other; p = 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 8.81, 95% CI 2-sided [4.58 to 13.03], Standard Error of Mean 2.14
Statistical Analysis 4: Comparison: A10 EZE (QM) vs A10 EvoMab QM; Test type: Superiority or Other; p = 0.006, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 8.28, 95% CI 2-sided [3.46 to 13.11], Standard Error of Mean 2.45
Statistical Analysis 5: Comparison: A80 PBO Q2W vs A80 EvoMab Q2W; Test type: Superiority or Other; p = 0.85, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 4.07, 95% CI 2-sided [-0.42 to 8.57], Standard Error of Mean 2.28
Statistical Analysis 6: Comparison: A80 PBO QM vs A80 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 7.05, 95% CI 2-sided [2.22 to 11.89], Standard Error of Mean 2.45
Statistical Analysis 7: Comparison: A80 EZE (Q2W) vs A80 EvoMab Q2W; Test type: Superiority or Other; p = 0.003, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 8.47, 95% CI 2-sided [4.07 to 12.87], Standard Error of Mean 2.23
Statistical Analysis 8: Comparison: A80 EZE (QM) vs A80 EvoMab QM; Test type: Superiority or Other; p = 0.003, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 7.14, 95% CI 2-sided [2.29 to 11.99], Standard Error of Mean 2.46
Statistical Analysis 9: Comparison: R5 PBO Q2W vs R5 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 3.20, 95% CI 2-sided [-1.33 to 7.73], Standard Error of Mean 2.30
Statistical Analysis 10: Comparison: R5 PBO QM vs R5 EvoMab QM; Test type: Superiority or Other; p = 0.010, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 7.35, 95% CI 2-sided [0.97 to 13.72], Standard Error of Mean 3.23
Statistical Analysis 11: Comparison: R40 PBO Q2W vs R40 EvoMab Q2W; Test type: Superiority or Other; p = 0.013, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 5.04, 95% CI 2-sided [0.52 to 9.56], Standard Error of Mean 2.29
Statistical Analysis 12: Comparison: R40 PBO QM vs R40 EvoMab QM; Test type: Superiority or Other; p = 0.002, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 4.84, 95% CI 2-sided [0.07 to 9.60], Standard Error of Mean 2.41
Statistical Analysis 13: Comparison: S40 PBO Q2W vs S40 EvoMab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 9.78, 95% CI 2-sided [4.05 to 15.51], Standard Error of Mean 2.90
Statistical Analysis 14: Comparison: S40 PBO QM vs S40 EvoMab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 9.06, 95% CI 2-sided [4.40 to 13.72], Standard Error of Mean 2.36

ADVERSE EVENTS:
Time Frame: From the first dose of blinded investigational product until the end of the study (up to 14 weeks).
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | A10 PBO Q2W | A10 PBO QM | A10 EZE (Q2W) | A10 EZE (QM) | A10 EvoMab Q2W | A10 EvoMab QM | A80 PBO Q2W | A80 PBO QM | A80 EZE (Q2W) | A80 EZE (QM) | A80 EvoMab Q2W | A80 EvoMab QM | R5 PBO Q2W | R5 PBO QM | R5 EvoMab Q2W | R5 EvoMab QM | R40 PBO Q2W | R40 PBO QM | R40 EvoMab Q2W | R40 EvoMab QM | S40 PBO Q2W | S40 PBO QM | S40 EvoMab Q2W | S40 EvoMab QM
Serious Adverse Events (participants affected / at risk) | 1/56 | 2/55 | 0/56 | 0/55 | 4/110 | 2/110 | 2/55 | 1/55 | 1/56 | 1/54 | 3/109 | 1/110 | 1/58 | 2/57 | 3/113 | 3/115 | 2/56 | 1/55 | 1/111 | 3/112 | 0/56 | 1/55 | 2/112 | 1/115
Other Adverse Events (participants affected / at risk) | 5/56 | 3/55 | 9/56 | 6/55 | 9/110 | 7/110 | 7/55 | 13/55 | 8/56 | 2/54 | 11/109 | 9/110 | 11/58 | 1/57 | 6/113 | 9/115 | 3/56 | 8/55 | 5/111 | 8/112 | 3/56 | 5/55 | 18/112 | 11/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A10 PBO Q2W (N=56) | A10 PBO QM (N=55) | A10 EZE (Q2W) (N=56) | A10 EZE (QM) (N=55) | A10 EvoMab Q2W (N=110) | A10 EvoMab QM (N=110) | A80 PBO Q2W (N=55) | A80 PBO QM (N=55) | A80 EZE (Q2W) (N=56) | A80 EZE (QM) (N=54) | A80 EvoMab Q2W (N=109) | A80 EvoMab QM (N=110) | R5 PBO Q2W (N=58) | R5 PBO QM (N=57) | R5 EvoMab Q2W (N=113) | R5 EvoMab QM (N=115) | R40 PBO Q2W (N=56) | R40 PBO QM (N=55) | R40 EvoMab Q2W (N=111) | R40 EvoMab QM (N=112) | S40 PBO Q2W (N=56) | S40 PBO QM (N=55) | S40 EvoMab Q2W (N=112) | S40 EvoMab QM (N=115)
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Campylobacter infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes simplex meningoencephalitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infected bites (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia mycoplasmal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleomorphic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coma (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Grand mal convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Affective disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glomerulonephritis acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hip arthroplasty (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aortic aneurysm (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peripheral artery stenosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | A10 PBO Q2W (N=56) | A10 PBO QM (N=55) | A10 EZE (Q2W) (N=56) | A10 EZE (QM) (N=55) | A10 EvoMab Q2W (N=110) | A10 EvoMab QM (N=110) | A80 PBO Q2W (N=55) | A80 PBO QM (N=55) | A80 EZE (Q2W) (N=56) | A80 EZE (QM) (N=54) | A80 EvoMab Q2W (N=109) | A80 EvoMab QM (N=110) | R5 PBO Q2W (N=58) | R5 PBO QM (N=57) | R5 EvoMab Q2W (N=113) | R5 EvoMab QM (N=115) | R40 PBO Q2W (N=56) | R40 PBO QM (N=55) | R40 EvoMab Q2W (N=111) | R40 EvoMab QM (N=112) | S40 PBO Q2W (N=56) | S40 PBO QM (N=55) | S40 EvoMab Q2W (N=112) | S40 EvoMab QM (N=115)
Constipation (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 4 | 1 | 0 | 4 | 2 | 0 | 1 | 0 | 2 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 1 | 2 | 1 | 2 | 2 | 2 | 1 | 3 | 0 | 4 | 0 | 1 | 2 | 0 | 5 | 2 | 1 | 0 | 1 | 6 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 3 | 4 | 1 | 2 | 3 | 0 | 2 | 1 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 3 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 2 | 0 | 0 | 1 | 0 | 3 | 1 | 1 | 1 | 2 | 1 | 0 | 0 | 2 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 3
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 3 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 1
Headache (Nervous system disorders) | 1 | 1 | 1 | 4 | 1 | 0 | 2 | 2 | 0 | 0 | 1 | 3 | 3 | 0 | 1 | 1 | 2 | 1 | 2 | 3 | 2 | 1 | 2 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.